CLINICAL TRIAL: NCT03858634
Title: KPL-716-C202: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Pilot Study to Investigate the Efficacy, Safety, and Tolerability of KPL-716 in Reducing Pruritus in Diseases Characterized by Chronic Pruritus
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of KPL-716 in Reducing Pruritus in Chronic Pruritic Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPL-716-C202; GX45045 (Other: Genentech, Inc.)
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Results first posted 2021-12-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Idiopathic Urticaria; Chronic Idiopathic Pruritus; Lichen Planus; Lichen Simplex Chronicus; Plaque Psoriasis
Keywords: pruritus, chronic pruritus, moderate to severe
MeSH Terms: conditions — Chronic Urticaria; Lichen Planus; Neurodermatitis; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KPL-716 (Experimental): Weekly for 8 weeks
  Interventions: Drug: KPL-716
- Placebo (Placebo Comparator): Weekly for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KPL-716 — A loading dose of KPL-716 720 mg (2x maintenance dose) administered via 2 subcutaneous (SC) injections within 30 minutes on Day 1. All subsequent doses of KPL-716 (360 mg maintenance dose) administered via a single SC injection.
  Other Names: Vixarelimab; RG6536
  Arms: KPL-716
Drug: Placebo — Placebo dose administered via 2 SC injections within 30 minutes on Day 1. All subsequent doses of placebo administered via a single SC injection.
  Arms: Placebo

SUMMARY:
Participants with diseases characterized by chronic pruritus experiencing moderate to severe pruritus will be enrolled in this pilot Phase 2 study.

The diseases characterized by chronic pruritus investigated in this pilot study currently include chronic idiopathic urticaria (CIU), chronic idiopathic pruritus (CIP), lichen planus (LP), lichen simplex chronicus (LSC) and plaque psoriasis (PPs).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years
2. Have clinical diagnosis of chronic idiopathic urticaria (CIU), chronic idiopathic pruritus (CIP), lichen planus (LP), lichen simplex chronicus (LSC) and plaque psoriasis (PPs) for at least 6 months
3. Moderate to severe pruritus
4. Female participants of childbearing potential must have a negative pregnancy test, be nonlactating, and have agreed to use a highly effective method of contraception, as specified in the protocol, from the Screening Visit until 10 weeks after final study drug administration
5. Able to comprehend and willing to sign an Informed Consent Form and able to abide by the study restrictions and comply with all study procedures for the duration of the study

Exclusion Criteria:

1. Use of prohibited medications within the indicated timeframe from Day 1 to the End of Study
2. Is currently using medication known to cause pruritus
3. Has any inflammatory, pruritic, and/or fibrotic skin condition other than the diagnosis that defines inclusion
4. Laboratory abnormalities that fall outside the windows specified in the protocol at the Screening Visit
5. Has an active infection, including skin infection
6. Any medical or psychiatric condition which, in the opinion of the Investigator or the Sponsor, may place the participant at increased risk as a result of study participation, interfere with study participation or study assessments, affect compliance with study requirements, or complicate interpretation of study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (14):
- United States (14):
  - Site 106, Anniston, Alabama
  - Site 110, Phoenix, Arizona
  - Site 114, Hot Springs, Arkansas
  - Site 103, Los Angeles, California
  - Site 113, Sweetwater, Florida
  - Site 105, Normal, Illinois
  - Site 112, Plainfield, Indiana
  - Site 119, New Orleans, Louisiana
  - Site 109, Fort Gratiot, Michigan
  - Site 123, New York, New York
  - Site 115, Johnston, Rhode Island
  - Site 104, Pflugerville, Texas
  - Site 101, San Antonio, Texas
  - Site 122, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study assigned participants to active treatment or placebo in 5 individual disease-specific cohorts: chronic idiopathic urticaria (CIU), chronic idiopathic pruritus (CIP), lichen planus (LP), lichen simplex chronicus (LSC) and plaque psoriasis (PPs). The participant flow data are presented by combined cohorts for public reporting purposes because the low numbers of participants in the individual disease-specific cohorts may cause re-identification concerns if presented separately.
Groups:
- KPL-716: KPL-716 weekly for 8 weeks
- Placebo: Placebo weekly for 8 weeks
Period: Overall Study
Arm/Group | KPL-716 | Placebo
Started | 39 | 19
Participants With Chronic Idiopathic Urticaria (CIU) | 4 | 2
Participants With Chronic Idiopathic Pruritus (CIP) | 14 | 9
Participants With Lichen Planus (LP) | 3 | 0
Participants With Lichen Simplex Chronicus (LSC) | 4 | 1
Participants With Plaque Psoriasis (PPs) | 14 | 7
Completed | 36 | 17
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other, Not Specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics data are presented by combined cohorts for public reporting purposes because the low numbers of participants in the individual disease-specific cohorts may cause re-identification concerns if presented separately.
Groups:
- Total: Total of all reporting groups
Arm/Group | KPL-716 | Placebo | Total
Number analyzed (Participants) | 39 | 19 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (11.51) | 53.3 (13.94) | 53.2 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 14 | 41
  Male | 12 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 14 | 48
  Black or African American | 4 | 4 | 8
  Asian | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 5 | 25
  Not Hispanic or Latino | 19 | 14 | 33
Weekly Average of Daily Worst Itch-Numeric Rating Scale (WI-NRS) [Mean (Standard Deviation); unit: score on a scale] — WI-NRS score: Participants were asked daily to assign a numerical score to the intensity of their most severe (worst) pruritus in the past 24 hours using a scale from 0 to 10, with 0 indicating no pruritus and 10 indicating the worst imaginable pruritus. Daily scores of Day -6 to Day 1 were averaged.
  score on a scale | 8.1 (0.93) | 8.3 (1.14) | 8.2 (1.00)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average WI-NRS at Week 8
Description: WI-NRS score: Participants were asked daily to assign a numerical score to the intensity of their most severe (worst) pruritus in the past 24 hours using a scale from 0 to 10, with 0 indicating no pruritus and 10 indicating the worst imaginable pruritus. Daily scores were averaged for a weekly score. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 8
Population: Modified intent to treat (mITT) set: all randomized participants who received at least 1 dose of KPL-716 or placebo and had at least 1 post-baseline efficacy assessment in the double-blind treatment period. Missing data were imputed using the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- KPL-716: CIU Cohort: Participants with CIU received KPL-716 weekly for 8 weeks
- Placebo: CIU Cohort: Participants with CIU received placebo weekly for 8 weeks
- KPL-716: CIP Cohort: Participants with CIP received KPL-716 weekly for 8 weeks
- Placebo: CIP Cohort: Participants with CIP received placebo weekly for 8 weeks
- KPL-716: LP Cohort: Participants with LP received KPL-716 weekly for 8 weeks
- Placebo: LP Cohort: Participants with LP received placebo weekly for 8 weeks
- KPL-716: LSC Cohort: Participants with LSC received KPL-716 weekly for 8 weeks
- Placebo: LSC Cohort: Participants with LSC received placebo weekly for 8 weeks
- KPL-716: PPs Cohort: Participants with PPs received KPL-716 weekly for 8 weeks
- Placebo: PPs Cohort: Participants with PPs received placebo weekly for 8 weeks
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
score on a scale | -4.3 (1.84) | -1.1 (2.66) | -4.3 (0.77) | -3.7 (0.96) | -3.1 (0.82) |  | -6.9 (0.81) | 0.7 (1.84) | -5.6 (0.69) | -2.5 (0.98)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Test type: Superiority; p = 0.3980, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; Least squares (LS) mean difference = -3.3, 80% CI 2-sided [-8.68 to 2.17], Standard Error of Mean 3.31
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Test type: Superiority; p = 0.6653, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -0.5, 80% CI 2-sided [-2.17 to 1.09], Standard Error of Mean 1.23
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Test type: Superiority; p = 0.0711, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -7.6, 80% CI 2-sided [-11.63 to -3.56], Standard Error of Mean 2.14
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Test type: Superiority; p = 0.0186, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -3.1, 80% CI 2-sided [-4.70 to -1.51], Standard Error of Mean 1.20

2. Secondary Outcome: Change From Baseline in Weekly Average WI-NRS Over Time
Description: as for outcome 1
Time Frame: Baseline, Weeks 1-18
Population: Modified intent to treat (mITT) set: all randomized participants who received at least 1 dose of KPL-716 or placebo and had at least 1 post-baseline efficacy assessment in the double-blind treatment period. Missing data were imputed using the last observation carried forward (LOCF) method. Once a participant started treatment period (through Week 8), missing data in treatment period were imputed. Once a participant started the follow up (FU) period, missing data in FU period were imputed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
score on a scale
  Change at Week 1 | -1.9 (0.59) | -0.9 (0.86) | -1.6 (0.55) | -1.4 (0.45) | -0.2 (0.13) |  | -3.0 (1.23) | -0.9 (NA) — 1 participant in this cohort. | -0.7 (0.17) | -0.2 (0.16)
  Change at Week 2 | -3.0 (0.79) | -1.3 (1.29) | -3.0 (0.60) | -2.9 (0.63) | -0.5 (0.58) |  | -4.0 (1.64) | -1.0 (NA) — 1 participant in this cohort. | -1.5 (0.27) | -0.7 (0.26)
  Change at Week 3 | -3.8 (1.25) | -1.6 (1.64) | -3.5 (0.61) | -2.4 (0.72) | -1.2 (0.99) |  | -4.6 (1.73) | -1.4 (NA) — 1 participant in this cohort. | -2.6 (0.39) | -0.9 (0.33)
  Change at Week 4 | -3.9 (1.59) | -1.5 (1.50) | -3.5 (0.64) | -3.0 (0.85) | -2.3 (1.78) |  | -5.0 (1.48) | -2.4 (NA) — 1 participant in this cohort. | -3.4 (0.48) | -1.2 (0.63)
  Change at Week 5 | -4.4 (1.83) | -1.6 (1.64) | -4.1 (0.73) | -3.1 (0.88) | -2.5 (1.91) |  | -5.4 (1.58) | -2.0 (NA) — 1 participant in this cohort. | -4.4 (0.65) | -1.5 (0.88)
  Change at Week 6 | -4.6 (1.72) | -1.8 (1.79) | -4.2 (0.74) | -3.7 (0.92) | -2.7 (1.90) |  | -5.8 (1.58) | -2.6 (NA) — 1 participant in this cohort. | -4.7 (0.65) | -1.6 (0.81)
  Change at Week 7 | -4.4 (1.75) | -2.6 (2.64) | -4.4 (0.77) | -3.7 (0.81) | -3.1 (1.94) |  | -6.3 (1.48) | -2.3 (NA) — 1 participant in this cohort. | -5.1 (0.69) | -1.9 (0.91)
  Change at Week 8 | -4.1 (1.84) | -1.6 (1.57) | -4.3 (0.75) | -3.7 (0.94) | -3.1 (1.94) |  | -6.0 (1.61) | -2.7 (NA) — 1 participant in this cohort. | -5.6 (0.66) | -2.5 (1.07)
  Change at Week 9: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 9 | -4.1 (1.73) | -1.6 (1.57) | -4.6 (0.88) | -3.8 (0.76) | -5.0 (1.00) |  | -6.0 (1.76) | -3.3 (NA) — 1 participant in this cohort. | -5.7 (0.70) | -2.5 (1.21)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 10 | -4.1 (1.69) | -2.2 (2.21) | -4.3 (0.87) | -4.7 (0.64) | -5.0 (1.00) |  | -6.3 (1.46) | -3.0 (NA) — 1 participant in this cohort. | -5.6 (0.75) | -2.2 (1.23)
  Change at Week 11: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 11 | -4.1 (1.74) | -2.2 (2.21) | -4.4 (0.90) | -4.9 (0.75) | -5.0 (1.00) |  | -6.3 (1.42) | -2.9 (NA) — 1 participant in this cohort. | -5.4 (0.78) | -2.2 (1.22)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 12 | -4.5 (1.72) | -2.2 (2.21) | -4.4 (0.86) | -4.3 (0.76) | -5.3 (0.71) |  | -6.5 (1.27) | -2.7 (NA) — 1 participant in this cohort. | -5.3 (0.80) | -2.2 (1.21)
  Change at Week 13: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 13 | -3.9 (1.85) | -2.2 (2.21) | -4.4 (0.83) | -4.2 (0.86) | -5.5 (0.50) |  | -6.6 (1.32) | -2.0 (NA) — 1 participant in this cohort. | -5.5 (0.83) | -2.3 (1.22)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 14 | -3.8 (1.75) | -2.2 (2.21) | -4.5 (0.80) | -4.1 (0.92) | -5.5 (0.50) |  | -6.4 (1.42) | -1.9 (NA) — 1 participant in this cohort. | -5.6 (0.81) | -2.3 (1.21)
  Change at Week 15: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 15 | -4.4 (1.68) | -2.2 (2.21) | -4.2 (0.85) | -3.8 (0.91) | -5.5 (0.50) |  | -6.8 (1.23) | -2.0 (NA) — 1 participant in this cohort. | -5.4 (0.86) | -2.6 (1.35)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 16 | -4.1 (1.74) | -2.2 (2.21) | -4.3 (0.87) | -3.5 (0.96) | -5.5 (0.50) |  | -6.6 (1.25) | -1.6 (NA) — 1 participant in this cohort. | -5.3 (0.86) | -2.6 (1.33)
  Change at Week 17: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 17 | -4.5 (1.81) | -2.2 (2.21) | -4.5 (0.89) | -3.4 (0.97) | -5.5 (0.50) |  | -6.8 (1.11) | -1.4 (NA) — 1 participant in this cohort. | -5.0 (0.99) | -2.7 (1.38)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 18 | -4.4 (1.67) | -2.2 (2.21) | -4.3 (0.97) | -3.4 (1.06) | -5.6 (0.57) |  | -6.9 (1.01) | -1.4 (NA) — 1 participant in this cohort. | -5.0 (1.01) | -2.7 (1.39)

3. Secondary Outcome: Percent Change From Baseline in Weekly Average WI-NRS Over Time
Description: as for outcome 1
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 1 | -23.5 (8.22) | -16.2 (11.84) | -19.5 (6.57) | -18.3 (8.20) | -2.4 (2.19) |  | -44.2 (12.54) | 16.9 (28.60) | -8.8 (1.84) | -3.4 (2.61)
  Change at Week 2 | -37.2 (12.11) | -20.6 (17.45) | -36.7 (7.42) | -36.5 (9.25) | -6.1 (4.37) |  | -59.8 (10.80) | 29.3 (24.62) | -17.8 (3.16) | -8.4 (4.46)
  Change at Week 3 | -46.9 (18.33) | -25.0 (26.41) | -43.4 (7.37) | -31.5 (9.19) | -15.0 (8.02) |  | -67.9 (12.89) | 25.9 (29.39) | -31.2 (4.14) | -11.2 (5.86)
  Change at Week 4 | -48.9 (19.96) | -20.0 (28.76) | -43.9 (7.92) | -38.4 (9.87) | -29.3 (18.23) |  | -71.7 (9.93) | 8.0 (22.65) | -41.7 (5.63) | -14.5 (7.96)
  Change at Week 5 | -54.7 (23.35) | -22.0 (33.65) | -51.6 (8.70) | -40.6 (10.84) | -31.1 (20.41) |  | -76.9 (13.08) | 13.8 (29.81) | -53.0 (7.11) | -17.7 (10.05)
  Change at Week 6 | -57.3 (21.58) | -23.8 (31.10) | -52.3 (9.11) | -47.9 (11.36) | -33.5 (17.50) |  | -81.5 (13.07) | 7.0 (29.80) | -56.5 (6.88) | -18.7 (9.72)
  Change at Week 7 | -53.6 (24.07) | -36.4 (34.67) | -54.3 (8.98) | -48.1 (11.19) | -39.4 (10.21) |  | -87.4 (11.02) | 7.8 (25.13) | -60.6 (7.48) | -22.5 (10.57)
  Change at Week 8 | -50.7 (21.56) | -19.0 (31.07) | -52.4 (9.32) | -48.8 (11.63) | -39.4 (10.21) |  | -85.0 (11.76) | 7.0 (26.80) | -66.5 (7.78) | -29.0 (11.00)
  Change at Week 9: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 9 | -51.1 (19.68) | -19.0 (28.35) | -55.7 (9.95) | -48.6 (11.50) | -62.5 (12.50) |  | -85.2 (14.00) | 4.0 (31.91) | -68.1 (8.42) | -28.5 (11.91)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 10 | -50.0 (20.26) | -27.9 (29.19) | -52.6 (9.40) | -58.7 (10.86) | -62.5 (12.50) |  | -86.8 (11.34) | -1.2 (25.85) | -67.0 (8.73) | -24.5 (12.35)
  Change at Week 11: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 11 | -50.4 (20.87) | -27.3 (30.07) | -52.8 (9.91) | -61.4 (11.45) | -62.5 (12.50) |  | -86.6 (10.72) | -0.4 (24.44) | -64.1 (8.66) | -24.8 (12.25)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 12 | -55.4 (21.36) | -28.2 (30.77) | -53.9 (9.88) | -53.2 (11.42) | -66.1 (8.93) |  | -89.0 (8.84) | -2.8 (20.15) | -62.2 (8.85) | -24.8 (12.52)
  Change at Week 13: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 13 | -47.2 (22.72) | -27.6 (32.73) | -53.8 (10.04) | -52.2 (11.59) | -68.8 (6.25) |  | -90.1 (10.04) | 6.1 (22.89) | -64.9 (9.22) | -25.2 (13.03)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 14 | -46.8 (20.94) | -27.7 (30.17) | -55.3 (10.15) | -51.4 (11.72) | -68.8 (6.25) |  | -88.8 (10.85) | 10.7 (24.74) | -65.9 (9.17) | -26.1 (12.97)
  Change at Week 15: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 15 | -53.6 (20.68) | -28.2 (29.79) | -50.8 (10.54) | -49.0 (12.18) | -68.8 (6.25) |  | -91.8 (9.58) | 3.0 (21.85) | -63.7 (9.87) | -29.5 (13.96)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 16 | -50.0 (21.31) | -28.0 (30.70) | -51.7 (10.86) | -44.7 (12.54) | -68.8 (6.25) |  | -90.6 (9.28) | 9.1 (21.17) | -62.7 (9.81) | -29.3 (13.88)
  Change at Week 17: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 17 | -55.0 (23.07) | -28.7 (33.24) | -54.2 (11.00) | -43.7 (12.70) | -68.8 (6.25) |  | -92.2 (8.10) | 6.8 (18.46) | -58.0 (11.35) | -30.8 (16.05)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 18 | -54.5 (20.93) | -28.9 (30.15) | -51.5 (12.05) | -43.7 (13.92) | -69.6 (7.14) |  | -92.1 (6.42) | 4.1 (14.63) | -58.1 (11.43) | -31.1 (16.17)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 1; Test type: Superiority; p = 0.6533, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -7.3, 80% CI 2-sided [-31.52 to 16.84], Standard Error of Mean 14.76
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 1; Test type: Superiority; p = 0.9077, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -1.2, 80% CI 2-sided [-15.16 to 12.69], Standard Error of Mean 10.51
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 1; Test type: Superiority; p = 0.2065, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -61.2, 80% CI 2-sided [-123.73 to 1.39], Standard Error of Mean 33.18
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 1; Test type: Superiority; p = 0.1133, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -5.3, 80% CI 2-sided [-9.56 to -1.07], Standard Error of Mean 3.19
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 2; Test type: Superiority; p = 0.4997, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -16.7, 80% CI 2-sided [-52.29 to 18.98], Standard Error of Mean 21.76
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 2; Test type: Superiority; p = 0.9919, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -0.1, 80% CI 2-sided [-15.83 to 15.59], Standard Error of Mean 11.85
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 2; Test type: Superiority; p = 0.0891, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -89.2, 80% CI 2-sided [-143.03 to -35.31], Standard Error of Mean 28.56
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 2; Test type: Superiority; p = 0.1029, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -9.4, 80% CI 2-sided [-16.67 to -2.12], Standard Error of Mean 5.47
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 3; Test type: Superiority; p = 0.5538, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -21.9, 80% CI 2-sided [-75.82 to 32.05], Standard Error of Mean 32.93
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 3; Test type: Superiority; p = 0.3252, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -11.9, 80% CI 2-sided [-27.51 to 3.73], Standard Error of Mean 11.78
Statistical Analysis 11: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 3; Test type: Superiority; p = 0.1106, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -93.8, 80% CI 2-sided [-158.11 to -29.52], Standard Error of Mean 34.10
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 3; Test type: Superiority; p = 0.0123, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -19.9, 80% CI 2-sided [-29.48 to -10.40], Standard Error of Mean 7.17
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.4791, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -28.9, 80% CI 2-sided [-87.63 to 29.81], Standard Error of Mean 35.86
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.6684, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -5.5, 80% CI 2-sided [-22.28 to 11.27], Standard Error of Mean 12.66
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.0937, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -79.7, 80% CI 2-sided [-129.22 to -30.13], Standard Error of Mean 26.28
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0120, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.2, 80% CI 2-sided [-40.21 to -14.27], Standard Error of Mean 9.75
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 5; Test type: Superiority; p = 0.4927, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -32.7, 80% CI 2-sided [-101.39 to 36.02], Standard Error of Mean 41.95
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 5; Test type: Superiority; p = 0.4409, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -10.9, 80% CI 2-sided [-29.35 to 7.49], Standard Error of Mean 13.90
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 5; Test type: Superiority; p = 0.1197, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -90.7, 80% CI 2-sided [-155.96 to -25.54], Standard Error of Mean 34.58
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 5; Test type: Superiority; p = 0.0102, ANOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -35.3, 80% CI 2-sided [-51.68 to -18.92], Standard Error of Mean 12.31
Statistical Analysis 21: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 6; Test type: Superiority; p = 0.4515, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -33.5, 80% CI 2-sided [-96.97 to 30.02], Standard Error of Mean 38.77
Statistical Analysis 22: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 6; Test type: Superiority; p = 0.7623, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -4.5, 80% CI 2-sided [-23.76 to 14.83], Standard Error of Mean 14.56
Statistical Analysis 23: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 6; Test type: Superiority; p = 0.1247, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -88.5, 80% CI 2-sided [-153.65 to -23.29], Standard Error of Mean 34.57
Statistical Analysis 24: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 6; Test type: Superiority; p = 0.0053, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -37.7, 80% CI 2-sided [-53.59 to -21.90], Standard Error of Mean 11.91
Statistical Analysis 25: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 7; Test type: Superiority; p = 0.7177, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -17.2, 80% CI 2-sided [-87.97 to 53.62], Standard Error of Mean 43.23
Statistical Analysis 26: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 7; Test type: Superiority; p = 0.6682, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -6.2, 80% CI 2-sided [-25.26 to 12.78], Standard Error of Mean 14.35
Statistical Analysis 27: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 7; Test type: Superiority; p = 0.0823, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -95.2, 80% CI 2-sided [-150.21 to -40.24], Standard Error of Mean 29.16
Statistical Analysis 28: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 7; Test type: Superiority; p = 0.0087, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -38.1, 80% CI 2-sided [-55.38 to -20.92], Standard Error of Mean 12.95
Statistical Analysis 29: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.4734, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -31.7, 80% CI 2-sided [-95.11 to 31.76], Standard Error of Mean 38.73
Statistical Analysis 30: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.8130, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -3.6, 80% CI 2-sided [-23.33 to 16.18], Standard Error of Mean 14.91
Statistical Analysis 31: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.0979, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -92.0, 80% CI 2-sided [-150.60 to -33.32], Standard Error of Mean 31.10
Statistical Analysis 32: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0122, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -37.5, 80% CI 2-sided [-55.48 to -19.61], Standard Error of Mean 13.48
Statistical Analysis 33: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 9; Test type: Superiority; p = 0.4310, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -32.1, 80% CI 2-sided [-89.98 to 25.81], Standard Error of Mean 35.35
Statistical Analysis 34: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 9; Test type: Superiority; p = 0.6452, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -7.1, 80% CI 2-sided [-27.38 to 13.12], Standard Error of Mean 15.22
Statistical Analysis 35: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 9; Test type: Superiority; p = 0.1375, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -89.2, 80% CI 2-sided [-159.04 to -19.44], Standard Error of Mean 37.02
Statistical Analysis 36: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 9; Test type: Superiority; p = 0.0143, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -39.6, 80% CI 2-sided [-58.97 to -20.15], Standard Error of Mean 14.59
Statistical Analysis 37: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 10; Test type: Superiority; p = 0.5867, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -22.1, 80% CI 2-sided [-81.70 to 37.52], Standard Error of Mean 36.40
Statistical Analysis 38: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 10; Test type: Superiority; p = 0.6745, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 6.1, 80% CI 2-sided [-12.99 to 25.27], Standard Error of Mean 14.38
Statistical Analysis 39: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 10; Test type: Superiority; p = 0.1039, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -85.6, 80% CI 2-sided [-142.18 to -29.09], Standard Error of Mean 29.99
Statistical Analysis 40: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 10; Test type: Superiority; p = 0.0116, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -42.5, 80% CI 2-sided [-62.60 to -22.36], Standard Error of Mean 15.12
Statistical Analysis 41: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 11; Test type: Superiority; p = 0.5807, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -23.1, 80% CI 2-sided [-84.55 to 38.26], Standard Error of Mean 37.49
Statistical Analysis 42: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 11; Test type: Superiority; p = 0.5765, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 8.6, 80% CI 2-sided [-11.55 to 28.80], Standard Error of Mean 15.16
Statistical Analysis 43: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 11; Test type: Superiority; p = 0.0933, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -86.2, 80% CI 2-sided [-139.70 to -32.75], Standard Error of Mean 28.36
Statistical Analysis 44: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 11; Test type: Superiority; p = 0.0173, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -39.3, 80% CI 2-sided [-59.29 to -19.37]
Statistical Analysis 45: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.5293, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.2, 80% CI 2-sided [-90.04 to 35.62], Standard Error of Mean 38.36
Statistical Analysis 46: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.9676, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -0.6, 80% CI 2-sided [-20.73 to 19.49], Standard Error of Mean 15.12
Statistical Analysis 47: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 12; Test type: Superiority; p = 0.0663, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -86.2, 80% CI 2-sided [-130.27 to -42.11], Standard Error of Mean 23.38
Statistical Analysis 48: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.0252, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -37.4, 80% CI 2-sided [-57.81 to -17.02], Standard Error of Mean 15.33
Statistical Analysis 49: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 13; Test type: Superiority; p = 0.6637, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -19.6, 80% CI 2-sided [-86.45 to 47.22], Standard Error of Mean 40.81
Statistical Analysis 50: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 13; Test type: Superiority; p = 0.9173, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -1.6, 80% CI 2-sided [-22.04 to 18.81], Standard Deviation 15.35
Statistical Analysis 51: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 13; Test type: Superiority; p = 0.0685, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -96.2, 80% CI 2-sided [-146.23 to -46.10], Standard Error of Mean 26.55
Statistical Analysis 52: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 13; Test type: Superiority; p = 0.0230, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -39.7, 80% CI 2-sided [-60.91 to -18.44], Standard Error of Mean 15.96
Statistical Analysis 53: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 14; Test type: Superiority; p = 0.6471, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -19.1, 80% CI 2-sided [-80.69 to 42.54], Standard Error of Mean 37.62
Statistical Analysis 54: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 14; Test type: Superiority; p = 0.8044, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -3.9, 80% CI 2-sided [-24.56 to 16.75], Standard Error of Mean 15.52
Statistical Analysis 55: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 14; Test type: Superiority; p = 0.0741, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -99.5, 80% CI 2-sided [-153.63 to -45.37], Standard Error of Mean 28.71
Statistical Analysis 56: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 14; Test type: Superiority; p = 0.0219, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -39.9, 80% CI 2-sided [-61.00 to -18.72], Standard Error of Mean 15.89
Statistical Analysis 57: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 15; Test type: Superiority; p = 0.5436, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -25.4, 80% CI 2-sided [-86.21 to 35.46], Standard Error of Mean 37.15
Statistical Analysis 58: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 15; Test type: Superiority; p = 0.9149, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -1.7, 80% CI 2-sided [-23.20 to 19.71], Standard Error of Mean 16.13
Statistical Analysis 59: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 15; Test type: Superiority; p = 0.0646, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -94.8, 80% CI 2-sided [-142.63 to -47.05], Standard Error of Mean 25.34
Statistical Analysis 60: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 15; Test type: Superiority; p = 0.0611, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -34.2, 80% CI 2-sided [-56.89 to -11.41], Standard Error of Mean 17.09
Statistical Analysis 61: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.6060, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -22.0, 80% CI 2-sided [-84.68 to 40.71], Standard Error of Mean 38.28
Statistical Analysis 62: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.6823, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -6.9, 80% CI 2-sided [-29.00 to 15.18], Standard Error of Mean 16.61
Statistical Analysis 63: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.0556, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -99.7, 80% CI 2-sided [-146.02 to -53.41], Standard Error of Mean 24.56
Statistical Analysis 64: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.0652, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -33.4, 80% CI 2-sided [-55.98 to -10.76], Standard Error of Mean 16.99
Statistical Analysis 65: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 17; Test type: Superiority; p = 0.5714, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -26.3, 80% CI 2-sided [-94.14 to 41.62], Standard Error of Mean 41.45
Statistical Analysis 66: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 17; Test type: Other; p = 0.5386, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -10.5, 80% CI 2-sided [-32.93 to 11.83], Standard Error of Mean 16.82
Statistical Analysis 67: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 17; Test type: Superiority; p = 0.0438, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -99.0, 80% CI 2-sided [-139.35 to -58.60], Standard Error of Mean 21.41
Statistical Analysis 68: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 17; Test type: Other; p = 0.1829, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.2, 80% CI 2-sided [-53.38 to -1.08], Standard Error of Mean 19.66
Statistical Analysis 69: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.5443, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -25.6, 80% CI 2-sided [-87.20 to 35.94], Standard Error of Mean 37.59
Statistical Analysis 70: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Superiority; p = 0.6748, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -7.9, 80% CI 2-sided [-32.39 to 16.66], Standard Error of Mean 18.43
Statistical Analysis 71: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.0297, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -96.2, 80% CI 2-sided [-128.19 to -64.19], Standard Error of Mean 16.97
Statistical Analysis 72: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Superiority; p = 0.1899, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.0, 80% CI 2-sided [-53.33 to -0.63], Standard Error of Mean 19.80

4. Secondary Outcome: Change From Baseline in Pruritus Visual Analog Scale (VAS) Over Time
Description: Participants were asked to place a line perpendicular to the VAS line at the point that represents the intensity of their average pruritus experienced over the previous 3 days using a scale from 0 to 10, with 0 indicating no pruritus and 10 indicating the worst imaginable pruritus.
Time Frame: Baseline, Weeks 1-8, 10, 12, 14, 16, 18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
units on a scale
  Change at Week 1 | -1.7 (0.98) | 0.0 (0.00) | -1.3 (0.79) | -2.0 (0.78) | -0.4 (0.26) |  | -4.0 (1.61) | -0.7 (NA) — 1 participant in this cohort | -1.3 (0.29) | -0.3 (0.28)
  Change at Week 2 | -2.8 (1.43) | 0.0 (0.00) | -3.0 (0.96) | -2.6 (0.62) | -0.4 (0.19) |  | -4.4 (1.80) | -1.0 (NA) — 1 participant in this cohort | -2.2 (0.55) | -0.7 (0.31)
  Change at Week 3 | -3.3 (1.52) | -0.1 (0.10) | -3.2 (1.09) | -3.4 (0.97) | -2.0 (1.36) |  | -5.2 (1.85) | -2.2 (NA) — 1 participant in this cohort | -3.4 (0.55) | -0.9 (0.81)
  Change at Week 4 | -4.3 (1.67) | 0.0 (0.00) | -3.7 (0.94) | -3.9 (0.95) | -2.8 (1.88) |  | -5.3 (1.66) | -2.2 (NA) — 1 participant in this cohort | -4.3 (0.54) | -1.4 (0.94)
  Change at Week 5 | -5.2 (1.82) | 0.0 (0.00) | -4.5 (1.01) | -4.7 (0.88) | -3.0 (1.86) |  | -5.7 (1.67) | -3.7 (NA) — 1 participant in this cohort | -4.3 (0.51) | -1.6 (0.99)
  Change at Week 6 | -4.4 (1.88) | 0.0 (0.00) | -4.5 (1.00) | -4.2 (1.07) | -3.1 (1.85) |  | -5.9 (1.57) | -2.0 (NA) — 1 participant in this cohort | -5.2 (0.54) | -1.9 (1.05)
  Change at Week 7 | -5.1 (1.78) | -0.1 (0.10) | -4.7 (1.05) | -4.7 (0.88) | -3.3 (1.85) |  | -6.1 (1.45) | -1.4 (NA) — 1 participant in this cohort | -5.3 (0.57) | -2.1 (1.27)
  Change at Week 8 | -4.2 (2.00) | 0.0 (0.00) | -4.4 (1.03) | -4.3 (0.95) | -3.3 (1.85) |  | -6.0 (1.42) | -1.8 (NA) — 1 participant in this cohort | -5.8 (0.61) | -2.2 (1.29)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 10 | -4.8 (1.86) | 0.0 (0.00) | -4.2 (1.07) | -5.8 (0.58) | -5.6 (0.85) |  | -6.2 (1.50) | -3.5 (NA) — 1 participant in this cohort | -5.9 (0.66) | -3.1 (1.36)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -4.1 (2.11) | 0.0 (0.00) | -4.7 (1.10) | -4.8 (1.18) | -5.1 (1.30) |  | -6.3 (1.37) | -3.5 (NA) — 1 participant in this cohort | -5.6 (0.71) | -3.8 (1.26)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 14 | -3.5 (2.19) | 0.0 (0.00) | -5.0 (1.00) | -4.2 (1.06) | -5.3 (1.10) |  | -6.4 (1.31) | -1.4 (NA) — 1 participant in this cohort | -5.8 (0.75) | -3.6 (1.37)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -4.5 (1.91) | -0.1 (0.05) | -4.2 (1.07) | -4.0 (1.13) | -5.6 (0.85) |  | -6.6 (1.12) | -0.8 (NA) — 1 participant in this cohort | -5.6 (0.79) | -3.5 (1.41)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -3.9 (2.07) | 0.0 (0.00) | -4.2 (1.22) | -3.6 (1.20) | -5.6 (2.40) |  | -7.0 (0.74) | -0.9 (NA) — 1 participant in this cohort | -5.4 (0.90) | -3.9 (1.31)

5. Secondary Outcome: Percent Change From Baseline in Pruritus VAS Over Time
Description: as for outcome 4
Time Frame: Baseline, Weeks 1-8, 10, 12, 14, 16, 18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 1 | -23.6 (13.76) | -8.3 (19.72) | -15.3 (9.17) | -24.8 (11.44) | -5.3 (1.80) |  | -76.1 (27.14) | 90.9 (85.95) | -15.4 (3.19) | -4.6 (4.52)
  Change at Week 2 | -37.4 (19.67) | -4.3 (28.19) | -34.2 (9.66) | -32.8 (12.04) | -5.1 (3.22) |  | -79.6 (34.28) | 81.3 (108.56) | -24.2 (5.50) | -10.1 (7.78)
  Change at Week 3 | -43.3 (19.79) | -2.6 (28.36) | -37.4 (12.12) | -44.5 (15.12) | -26.2 (8.32) |  | -97.1 (28.92) | 96.7 (91.57) | -40.6 (6.26) | -10.3 (8.87)
  Change at Week 4 | -54.9 (19.93) | -0.9 (28.57) | -44.4 (10.57) | -50.7 (13.18) | -37.3 (12.60) |  | -93.6 (28.13) | 74.8 (89.08) | -52.7 (6.55) | -16.0 (9.27)
  Change at Week 5 | -66.3 (21.37) | -0.2 (30.63) | -54.1 (10.84) | -60.4 (13.52) | -40.0 (15.97) |  | -99.4 (26.68) | 64.0 (84.47) | -52.5 (6.54) | -19.1 (9.26)
  Change at Week 6 | -57.2 (22.58) | -1.2 (32.37) | -53.0 (11.31) | -52.4 (14.11) | -41.6 (17.99) |  | -101.0 (24.68) | 76.3 (78.14) | -63.5 (6.90) | -21.5 (9.77)
  Change at Week 7 | -65.7 (18.99) | 0.1 (27.22) | -55.7 (10.97) | -60.8 (13.68) | -44.3 (21.36) |  | -101.8 (22.55) | 73.6 (71.40) | -64.6 (7.89) | -25.4 (11.18)
  Change at Week 8 | -54.1 (22.59) | -0.4 (32.38) | -52.1 (11.11) | -55.0 (13.86) | -44.3 (21.36) |  | -99.2 (23.11) | 63.8 (73.18) | -70.9 (8.44) | -25.2 (11.96)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 10 | -61.6 (20.31) | 0.7 (29.11) | -50.7 (10.73) | -72.2 (12.39) | -76.9 (0.00) |  | -103.9 (22.62) | 57.5 (71.64) | -70.6 (8.32) | -36.2 (12.71)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -51.9 (21.21) | 3.3 (30.40) | -56.3 (12.44) | -58.7 (14.37) | -69.7 (0.00) |  | -102.9 (21.13) | 46.3 (66.92) | -67.6 (8.32) | -45.5 (12.71)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 14 | -44.2 (20.40) | 4.4 (29.24) | -60.8 (11.32) | -51.2 (13.07) | -72.9 (0.00) |  | -103.3 (19.74) | 64.5 (62.52) | -69.6 (8.91) | -42.5 (13.61)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -56.8 (14.02) | 5.1 (20.09) | -49.5 (11.91) | -48.9 (13.75) | -76.9 (0.00) |  | -102.0 (16.87) | 57.2 (53.41) | -68.1 (9.43) | -41.6 (14.40)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -47.8 (14.97) | 6.8 (21.45) | -49.1 (13.66) | -45.0 (15.77) | -74.6 (0.00) |  | -101.3 (9.93) | 29.5 (31.43) | -64.5 (10.23) | -46.0 (15.63)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 1; Test type: Superiority; p = 0.5763, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -15.3, 80% CI 2-sided [-55.37 to 24.78], Standard Error of Mean 24.47
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 1; Test type: Superiority; p = 0.5214, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 9.6, 80% CI 2-sided [-9.86 to 29.01], Standard Error of Mean 14.66
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 1; Test type: Superiority; p = 0.2536, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -167.0, 80% CI 2-sided [-365.51 to 31.54], Standard Error of Mean 105.28
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 1; Test type: Superiority; p = 0.0670, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -10.8, 80% CI 2-sided [-18.20 to -3.44], Standard Error of Mean 5.55
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 2; Test type: Superiority; p = 0.4133, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -33.1, 80% CI 2-sided [-90.43 to 24.15], Standard Error of Mean 34.98
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 2; Test type: Superiority; p = 0.9305, ANCOVA; LS mean difference = -1.4, 80% CI 2-sided [-21.83 to 19.11], Standard Error of Mean 15.44
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 2; Test type: Superiority; p = 0.3499, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -160.9, 80% CI 2-sided [-411.65 to 89.86], Standard Error of Mean 132.98
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 2; Test type: Superiority; p = 0.1588, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -14.0, 80% CI 2-sided [-26.74 to -1.33], Standard Error of Mean 9.55
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 3; Test type: Superiority; p = 0.3319, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -40.6, 80% CI 2-sided [-98.26 to 17.00], Standard Error of Mean 35.19
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 3; Test type: Superiority; p = 0.7179, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 7.1, 80% CI 2-sided [-18.59 to 32.80], Standard Error of Mean 19.39
Statistical Analysis 11: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 3; Test type: Superiority; p = 0.2261, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -193.8, 80% CI 2-sided [-405.34 to 17.67], Standard Error of Mean 112.17
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 3; Test type: Superiority; p = 0.0123, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -30.3, 80% CI 2-sided [-44.75 to -15.80], Standard Error of Mean 10.88
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.2253, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -54.0, 80% CI 2-sided [-112.02 to 4.09], Standard Error of Mean 35.45
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.7149, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 6.3, 80% CI 2-sided [-16.14 to 28.66], Standard Error of Mean 16.90
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.2627, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -168.4, 80% CI 2-sided [-374.16 to 37.36], Standard Error of Mean 109.12
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0047, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -36.7, 80% CI 2-sided [-51.87 to -21.60], Standard Error of Mean 11.38
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 5; Test type: Superiority; p = 0.1803, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -66.1, 80% CI 2-sided [-128.37 to -3.88], Standard Error of Mean 38.01
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 5; Test type: Superiority; p = 0.7174, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 6.4, 80% CI 2-sided [-16.62 to 29.35], Standard Error of Mean 17.34
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 5; Test type: Superiority; p = 0.2551, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -163.4, 80% CI 2-sided [-358.51 to 31.72], Standard Error of Mean 103.47
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 5; Test type: Superiority; p = 0.0086, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -33.5, 80% CI 2-sided [-48.58 to -18.36], Standard Error of Mean 11.36
Statistical Analysis 21: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 6; Test type: Superiority; p = 0.2576, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -56.0, 80% CI 2-sided [-121.78 to 9.78], Standard Error of Mean 40.16
Statistical Analysis 22: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 6; Test type: Superiority; p = 0.9722, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -0.6, 80% CI 2-sided [-24.62 to 23.34], Standard Error of Mean 18.09
Statistical Analysis 23: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 6; Test type: Superiority; p = 0.2051, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -177.4, 80% CI 2-sided [-357.85 to 3.13], Standard Error of Mean 95.72
Statistical Analysis 24: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 6; Test type: Superiority; p = 0.0025, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -42.0, 80% CI 2-sided [-57.98 to -26.08], Standard Error of Mean 11.99
Statistical Analysis 25: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 7; Test type: Superiority; p = 0.1465, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -65.8, 80% CI 2-sided [-121.14 to -10.50], Standard Error of Mean 33.78
Statistical Analysis 26: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 7; Test type: Superiority; p = 0.7734, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 5.1, 80% CI 2-sided [-18.13 to 28.37], Standard Error of Mean 17.54
Statistical Analysis 27: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 7; Test type: Superiority; p = 0.1826, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -175.5, 80% CI 2-sided [-340.37 to -10.56], Standard Error of Mean 87.45
Statistical Analysis 28: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 7; Test type: Superiority; p = 0.0105, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -39.2, 80% CI 2-sided [-57.40 to -20.93], Standard Error of Mean 13.71
Statistical Analysis 29: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.2737, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -53.7, 80% CI 2-sided [-119.49 to 12.09], Standard Error of Mean 40.17
Statistical Analysis 30: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.8692, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 3.0, 80% CI 2-sided [-20.59 to 26.52], Standard Error of Mean 17.77
Statistical Analysis 31: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.2106, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -163.0, 80% CI 2-sided [-332.06 to 5.99], Standard Error of Mean 89.64
Statistical Analysis 32: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0060, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -45.7, 80% CI 2-sided [-65.19 to -26.14], Standard Error of Mean 14.67
Statistical Analysis 33: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 10; Test type: Superiority; p = 0.1831, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -62.3, 80% CI 2-sided [-121.44 to -3.13], Standard Error of Mean 36.12
Statistical Analysis 34: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 10; Test type: Superiority; p = 0.2061, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 21.5, 80% CI 2-sided [-0.31 to 43.30], Standard Error of Mean 16.39
Statistical Analysis 35: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 10; Test type: Superiority; p = 0.2073, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -161.4, 80% CI 2-sided [-326.83 to 4.12], Standard Error of Mean 87.75
Statistical Analysis 36: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 10; Test type: Superiority; p = 0.0371, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -34.4, 80% CI 2-sided [-54.62 to -14.10], Standard Error of Mean 15.19
Statistical Analysis 37: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.2393, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -55.2, 80% CI 2-sided [-117.01 to 6.54], Standard Error of Mean 37.72
Statistical Analysis 38: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.9019, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 2.4, 80% CI 2-sided [-22.91 to 27.67], Standard Error of Mean 19.01
Statistical Analysis 39: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 12; Test type: Superiority; p = 0.2103, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -149.2, 80% CI 2-sided [-303.77 to 5.35], Standard Error of Mean 81.97
Statistical Analysis 40: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.1634, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -22.1, 80% CI 2-sided [-42.40 to -1.88], Standard Error of Mean 15.20
Statistical Analysis 41: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 14; Test type: Superiority; p = 0.2727, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -48.6, 80% CI 2-sided [-108.04 to 10.80], Standard Error of Mean 36.28
Statistical Analysis 42: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 14; Test type: Superiority; p = 0.5839, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -9.6, 80% CI 2-sided [-32.65 to 13.36], Standard Error of Mean 17.29
Statistical Analysis 43: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 14; Test type: Superiority; p = 0.1597, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -167.8, 80% CI 2-sided [-312.25 to -23.45], Standard Error of Mean 76.58
Statistical Analysis 44: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 14; Test type: Superiority; p = 0.1138, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.1, 80% CI 2-sided [-48.81 to -5.43], Standard Error of Mean 16.27
Statistical Analysis 45: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.0888, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -62.0, 80% CI 2-sided [-102.78 to -21.13], Standard Error of Mean 24.93
Statistical Analysis 46: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.9741, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -0.6, 80% CI 2-sided [-24.79 to 23.60], Standard Error of Mean 18.19
Statistical Analysis 47: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.1354, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -159.2, 80% CI 2-sided [-282.59 to -35.87], Standard Error of Mean 65.42
Statistical Analysis 48: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.1425, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -26.5, 80% CI 2-sided [-49.41 to -3.52], Standard Error of Mean 17.21
Statistical Analysis 49: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.1326, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -54.6, 80% CI 2-sided [-98.18 to -11.01], Standard Error of Mean 26.61
Statistical Analysis 50: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Other; p = 0.8433, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -4.2, 80% CI 2-sided [-31.95 to 23.58], Standard Error of Mean 20.87
Statistical Analysis 51: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.0768, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -130.8, 80% CI 2-sided [-203.39 to -58.19], Standard Error of Mean 38.50
Statistical Analysis 52: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Superiority; p = 0.3341, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -18.6, 80% CI 2-sided [-43.49 to 6.34], Standard Error of Mean 18.69

6. Secondary Outcome: Change From Baseline in 5-D Pruritus Total Score Over Time
Description: This tool evaluates pruritus in 5 domains: duration, degree, direction, disability and distribution. Duration, degree and direction each consist of 1 item. The disability domain contains 4 items and the distribution domain includes 16 items. The first 4 domains are measured on a 5-point Likert scale. The scores from each domain are added together to obtain a total 5-D score ranging from 5 (no pruritus) and 25 (most severe pruritus).
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
units on a scale
  Change at Week 2 | -6.3 (2.78) | 0.0 (0.00) | -4.4 (1.06) | -4.0 (1.35) | -2.3 (1.20) |  | -6.8 (2.10) | -4.0 (NA) — 1 participant in this cohort. | -5.0 (1.19) | -3.6 (1.29)
  Change at Week 4 | -8.5 (2.02) | 0.5 (0.50) | -4.5 (1.27) | -5.4 (1.65) | -7.3 (4.06) |  | -7.3 (2.78) | -4.0 (NA) — 1 participant in this cohort. | -7.7 (1.05) | -4.1 (1.81)
  Change at Week 6 | -8.3 (2.17) | 0.5 (0.50) | -6.6 (1.23) | -5.8 (1.47) | -8.0 (4.16) |  | -8.5 (2.90) | -7.0 (NA) — 1 participant in this cohort. | -8.2 (1.05) | -5.0 (1.79)
  Change at Week 8 | -7.5 (2.22) | -0.5 (0.50) | -6.5 (1.32) | -6.8 (1.23) | -8.0 (4.16) |  | -8.8 (2.95) | -7.0 (NA) — 1 participant in this cohort. | -9.4 (1.09) | -5.0 (1.75)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 10 | -8.0 (1.68) | -1.0 (1.00) | -6.6 (1.50) | -7.9 (0.63) | -12.0 (2.00) |  | -9.5 (2.87) | -7.0 (NA) — 1 participant in this cohort. | -9.4 (1.46) | -6.0 (1.81)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -7.0 (2.42) | 0.0 (0.00) | -6.3 (1.33) | -6.3 (1.04) | -12.0 (2.00) |  | -9.8 (2.63) | -8.0 (NA) — 1 participant in this cohort. | -9.6 (1.32) | -6.3 (1.71)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 14 | -4.0 (3.37) | 0.0 (0.00) | -6.7 (1.08) | -6.1 (1.17) | -12.0 (2.00) |  | -9.5 (2.87) | -4.0 (NA) — 1 participant in this cohort. | -9.6 (1.53) | -6.5 (1.78)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -7.8 (2.10) | 0.5 (0.50) | -7.1 (1.77) | -5.0 (1.47) | -11.5 (2.50) |  | -10.0 (2.38) | -2.0 (NA) — 1 participant in this cohort. | -9.6 (1.48) | -7.2 (1.97)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -6.5 (2.50) | 0.5 (0.50) | -6.3 (1.82) | -4.6 (1.42) | -13.5 (3.50) |  | -10.0 (2.38) | -2.0 (NA) — 1 participant in this cohort. | -8.9 (1.57) | -7.0 (1.65)

7. Secondary Outcome: Percent Change From Baseline in 5-D Pruritus Total Score Over Time
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 2 | -31.3 (13.40) | 0.0 (18.98) | -24.2 (6.00) | -20.6 (7.48) | -11.8 (8.46) |  | -44.0 (3.43) | 8.4 (8.04) | -25.4 (5.38) | -18.8 (7.61)
  Change at Week 4 | -42.7 (9.40) | 2.4 (13.31) | -24.1 (7.03) | -29.2 (8.77) | -35.1 (12.38) |  | -49.1 (2.09) | 23.0 (4.90) | -40.3 (5.55) | -20.8 (7.85)
  Change at Week 6 | -41.4 (10.22) | 2.3 (14.48) | -35.9 (6.66) | -31.6 (8.31) | -38.8 (17.46) |  | -56.5 (1.49) | 9.1 (3.49) | -43.3 (5.67) | -25.9 (8.02)
  Change at Week 8 | -37.7 (10.85) | -2.2 (15.36) | -34.4 (6.30) | -37.2 (7.85) | -38.8 (17.46) |  | -58.1 (0.83) | 10.1 (1.95) | -49.1 (5.49) | -25.7 (7.77)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 10 | -40.1 (8.46) | -4.5 (11.98) | -35.2 (6.47) | -43.1 (7.48) | -58.2 (0.00) |  | -62.1 (3.76) | 6.6 (8.82) | -49.1 (6.55) | -29.6 (10.06)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -33.3 (9.21) | -0.8 (13.05) | -33.5 (6.64) | -34.4 (7.66) | -58.2 (0.00) |  | -62.8 (3.53) | -3.4 (8.28) | -50.2 (5.86) | -31.4 (9.00)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 14 | -17.9 (14.08) | -1.1 (19.95) | -36.2 (5.83) | -33.3 (6.74) | -58.2 (0.00) |  | -62.1 (3.76) | 20.2 (8.82) | -49.7 (7.04) | -33.1 (10.81)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -37.7 (8.29) | 1.7 (11.74) | -37.0 (8.29) | -27.8 (9.57) | -55.4 (0.00) |  | -63.6 (3.33) | 18.5 (7.81) | -49.9 (7.08) | -36.8 (10.88)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -31.3 (10.41) | 1.6 (14.75) | -32.9 (8.83) | -25.0 (10.19) | -64.7 (0.00) |  | -63.6 (3.33) | 18.5 (7.81) | -46.6 (7.43) | -35.5 (11.41)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 2; Test type: Superiority; p = 0.4995, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -40.9, 80% CI 2-sided [-166.52 to 84.74], Standard Error of Mean 40.82
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 2; Test type: Superiority; p = 0.7071, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -3.7, 80% CI 2-sided [-16.37 to 9.06], Standard Error of Mean 9.59
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 2; Test type: Superiority; p = 0.0305, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -52.5, 80% CI 2-sided [-70.18 to -34.77], Standard Error of Mean 9.39
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 2; Test type: Superiority; p = 0.4884, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -6.6, 80% CI 2-sided [-19.01 to 5.81], Standard Error of Mean 9.33
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.2885, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -45.3, 80% CI 2-sided [-104.93 to 14.35], Standard Error of Mean 31.63
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.6505, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 5.2, 80% CI 2-sided [-9.73 to 20.06], Standard Error of Mean 11.24
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.0062, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -72.1, 80% CI 2-sided [-82.91 to -61.34], Standard Error of Mean 5.72
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0571, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -19.6, 80% CI 2-sided [-32.34 to -6.76], Standard Error of Mean 9.62
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 6; Test type: Superiority; LS mean difference = -50.1, Standard Error of Mean 0.00
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 6; Test type: Superiority; p = 0.6927, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -4.3, 80% CI 2-sided [-18.38 to 9.84], Standard Error of Mean 10.65
Statistical Analysis 11: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 6; Test type: Superiority; p = 0.0038, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -65.6, 80% CI 2-sided [-73.33 to -57.94], Standard Error of Mean 4.08
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 6; Test type: Superiority; p = 0.0940, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -17.4, 80% CI 2-sided [-30.43 to -4.30], Standard Error of Mean 9.82
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.1694, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -72.4, 80% CI 2-sided [-133.10 to -11.65], Standard Error of Mean 19.73
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.7811, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 2.8, 80% CI 2-sided [-10.50 to 16.18], Standard Error of Mean 10.07
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.0011, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -68.2, 80% CI 2-sided [-72.51 to -63.91], Standard Error of Mean 2.28
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0245, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -23.4, 80% CI 2-sided [-36.02 to -10.70], Standard Error of Mean 9.52
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 10; Test type: Superiority; p = 0.0603, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -61.8, 80% CI 2-sided [-79.88 to -43.74], Standard Error of Mean 5.87
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 10; Test type: Superiority; p = 0.4365, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 7.9, 80% CI 2-sided [-5.29 to 21.04], Standard Error of Mean 9.89
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 10; Test type: Superiority; p = 0.0218, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -68.7, 80% CI 2-sided [-88.11 to -49.26], Standard Error of Mean 10.30
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 10; Test type: Superiority; p = 0.1238, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -19.5, 80% CI 2-sided [-35.65 to -3.45], Standard Error of Mean 12.07
Statistical Analysis 21: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.1437, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -54.8, 80% CI 2-sided [-98.88 to -10.72], Standard Error of Mean 23.38
Statistical Analysis 22: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.9279, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 0.9, 80% CI 2-sided [-12.56 to 14.43], Standard Error of Mean 10.14
Statistical Analysis 23: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 12; Test type: Superiority; p = 0.0254, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -59.5, 80% CI 2-sided [-77.69 to -41.24], Standard Error of Mean 9.67
Statistical Analysis 24: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.0994, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -18.8, 80% CI 2-sided [-33.23 to -4.43], Standard Error of Mean 10.80
Statistical Analysis 25: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 14; Test type: Superiority; p = 0.3656, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -45.7, 80% CI 2-sided [-119.90 to 28.54], Standard Error of Mean 39.36
Statistical Analysis 26: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 14; Test type: Superiority; p = 0.7465, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -2.9, 80% CI 2-sided [-14.79 to 8.94], Standard Error of Mean 8.92
Statistical Analysis 27: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 14; Test type: Superiority; p = 0.0153, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -82.3, 80% CI 2-sided [-101.75 to -62.90], Standard Error of Mean 10.30
Statistical Analysis 28: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 14; Test type: Superiority; p = 0.2184, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -16.6, 80% CI 2-sided [-33.88 to 0.72], Standard Error of Mean 12.97
Statistical Analysis 29: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.7726, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -8.1, 80% CI 2-sided [-50.37 to 34.07], Standard Error of Mean 25.78
Statistical Analysis 30: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.4760, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -9.2, 80% CI 2-sided [-26.07 to 7.63], Standard Error of Mean 12.66
Statistical Analysis 31: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.0121, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -82.1, 80% CI 2-sided [-99.26 to -64.87], Standard Error of Mean 9.12
Statistical Analysis 32: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.3329, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -13.0, 80% CI 2-sided [-30.43 to 4.40], Standard Error of Mean 13.06
Statistical Analysis 33: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.9564, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -1.7, 80% CI 2-sided [-48.31 to 44.92], Standard Error of Mean 28.46
Statistical Analysis 34: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Superiority; p = 0.5661, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -7.9, 80% CI 2-sided [-25.84 to 10.06], Standard Error of Mean 13.49
Statistical Analysis 35: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.0121, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -82.1, 80% CI 2-sided [-99.26 to -64.87], Standard Error of Mean 9.12
Statistical Analysis 36: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Superiority; p = 0.4275, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -11.1, 80% CI 2-sided [-29.40 to 7.13], Standard Error of Mean 13.70

8. Secondary Outcome: Percentage of Participants Achieving ≥4-Point Reduction From Baseline in Weekly Average WI-NRS Over Time
Description: as for outcome 1
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percentage of participants
  Change at Week 1 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 84.2] | 21.4 [4.7 to 50.8] | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 70.8] |  | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 41.0]
  Change at Week 2 | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 28.6 [8.4 to 58.1] | 33.3 [7.5 to 70.1] | 0.0 [0.0 to 70.8] |  | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 41.0]
  Change at Week 3 | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 42.9 [17.7 to 71.1] | 33.3 [7.5 to 70.1] | 0.0 [0.0 to 70.8] |  | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 97.5] | 21.4 [4.7 to 50.8] | 0.0 [0.0 to 41.0]
  Change at Week 4 | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 42.9 [17.7 to 71.1] | 44.4 [13.7 to 78.8] | 33.3 [0.8 to 90.6] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 42.9 [17.7 to 71.1] | 14.3 [0.4 to 57.9]
  Change at Week 5 | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 50.0 [23.0 to 77.0] | 44.4 [13.7 to 78.8] | 33.3 [0.8 to 90.6] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 50.0 [23.0 to 77.0] | 14.3 [0.4 to 57.9]
  Change at Week 6 | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 57.1 [28.9 to 82.3] | 66.7 [29.9 to 92.5] | 33.3 [0.8 to 90.6] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 57.1 [28.9 to 82.3] | 14.3 [0.4 to 57.9]
  Change at Week 7 | 50.0 [6.8 to 93.2] | 50.0 [1.3 to 98.7] | 57.1 [28.9 to 82.3] | 55.6 [21.2 to 86.3] | 66.7 [9.4 to 99.2] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 64.3 [35.1 to 87.2] | 14.3 [0.4 to 57.9]
  Change at Week 8 | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 57.1 [28.9 to 82.3] | 66.7 [29.9 to 92.5] | 66.7 [9.4 to 99.2] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 71.4 [41.9 to 91.6] | 28.6 [3.7 to 71.0]
  Change at Week 9: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 9 | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 58.3 [27.7 to 84.8] | 55.6 [21.2 to 86.3] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 78.6 [49.2 to 95.3] | 28.6 [3.7 to 71.0]
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 10 | 25.0 [0.6 to 80.6] | 50.0 [1.3 to 98.7] | 50.0 [21.1 to 78.9] | 77.8 [40.0 to 97.2] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 78.6 [49.2 to 95.3] | 14.3 [0.4 to 57.9]
  Change at Week 11: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 11 | 50.0 [6.8 to 93.2] | 50.0 [1.3 to 98.7] | 58.3 [27.7 to 84.8] | 77.8 [40.0 to 97.2] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 64.3 [35.1 to 87.2] | 14.3 [0.4 to 57.9]
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 12 | 50.0 [6.8 to 93.2] | 50.0 [1.3 to 98.7] | 58.3 [27.7 to 84.8] | 66.7 [29.9 to 92.5] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 64.3 [35.1 to 87.2] | 14.3 [0.4 to 57.9]
  Change at Week 13: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 13 | 25.0 [0.6 to 80.6] | 50.0 [1.3 to 98.7] | 58.3 [27.7 to 84.8] | 55.6 [21.2 to 86.3] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 71.4 [41.9 to 91.6] | 14.3 [0.4 to 57.9]
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 14 | 25.0 [0.6 to 80.6] | 50.0 [1.3 to 98.7] | 58.3 [27.7 to 84.8] | 55.6 [21.2 to 86.3] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 71.4 [41.9 to 91.6] | 14.3 [0.4 to 57.9]
  Change at Week 15: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 15 | 50.0 [6.8 to 93.2] | 50.0 [1.3 to 98.7] | 50.0 [21.1 to 78.9] | 44.4 [13.7 to 78.8] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 71.4 [41.9 to 91.6] | 28.6 [3.7 to 71.0]
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 16 | 25.0 [0.6 to 80.6] | 50.0 [1.3 to 98.7] | 58.3 [27.7 to 84.8] | 44.4 [13.7 to 78.8] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 71.4 [41.9 to 91.6] | 28.6 [3.7 to 71.0]
  Change at Week 17: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 17 | 75.0 [19.4 to 99.4] | 50.0 [1.3 to 98.7] | 50.0 [21.1 to 78.9] | 44.4 [13.7 to 78.8] | 100.0 [15.8 to 100.0] |  | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 97.5] | 71.4 [41.9 to 91.6] | 28.6 [3.7 to 71.0]
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 14 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 18 | 75.0 [19.4 to 99.4] | 50.0 [1.3 to 98.7] | 58.3 [27.7 to 84.8] | 44.4 [13.7 to 78.8] | 100.0 [15.8 to 100.0] |  | 100.0 [39.8 to 100.0] | 0.0 [0.0 to 97.5] | 71.4 [41.9 to 91.6] | 28.6 [3.7 to 71.0]

9. Secondary Outcome: Change From Baseline in Weekly Average Itch Severity Score: CIU Cohort Only
Description: Participants were asked daily to self-assess the intensity of their pruritus on a Weekly Average Itch Severity Score, which is a Component of Urticaria Activity Score 7 (UAS7). The score for pruritis was graded from 0 (none) to 3 (intense), which was averaged over 7 consecutive days. The greater the severity of the disease the higher the score. Per protocol, the UAS7 tool was completed only by participants in the CIU Cohort.
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort
Number analyzed (Participants) | 4 | 2
score on a scale
  Change at Week 1 | -0.7 (0.13) | 0.3 (0.29)
  Change at Week 2 | -0.9 (0.15) | -0.2 (0.21)
  Change at Week 3 | -1.0 (0.36) | -0.4 (0.36)
  Change at Week 4 | -1.2 (0.30) | -0.2 (0.21)
  Change at Week 5 | -1.2 (0.28) | -0.2 (0.21)
  Change at Week 6 | -1.4 (0.22) | -0.1 (0.14)
  Change at Week 7 | -1.1 (0.30) | -0.4 (0.43)
  Change at Week 8 | -0.8 (0.40) | -0.1 (0.14)
  Change at Week 9 | -1.2 (0.27) | -0.1 (0.14)
  Change at Week 10 | -1.1 (0.35) | -0.5 (0.50)
  Change at Week 11 | -1.0 (0.39) | -0.6 (0.57)
  Change at Week 12 | -1.0 (0.39) | -0.6 (0.57)
  Change at Week 13 | -0.7 (0.44) | -0.6 (0.57)
  Change at Week 14 | -0.9 (0.41) | -0.6 (0.57)
  Change at Week 15 | -1.1 (0.38) | -0.6 (0.57)
  Change at Week 16 | -0.9 (0.39) | -0.6 (0.57)
  Change at Week 17 | -1.1 (0.35) | -0.6 (0.57)
  Change at Week 18 | -1.3 (0.24) | -0.6 (0.57)

10. Secondary Outcome: Percent Change From Baseline in Weekly Average Itch Severity Score: CIU Cohort Only
Description: as for outcome 9
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort
Number analyzed (Participants) | 4 | 2
percent change
  Change at Week 1 | -26.6 (5.36) | -13.3 (13.33)
  Change at Week 2 | -36.4 (4.94) | -10.0 (10.00)
  Change at Week 3 | -40.8 (11.29) | -16.7 (16.67)
  Change at Week 4 | -45.5 (8.82) | -10.0 (10.00)
  Change at Week 5 | -48.7 (8.76) | -10.0 (10.00)
  Change at Week 6 | -54.6 (5.27) | -6.7 (6.67)
  Change at Week 7 | -43.8 (8.48) | -20.0 (20.00)
  Change at Week 8 | -31.5 (12.83) | -6.7 (6.67)
  Change at Week 9 | -48.3 (6.99) | -6.7 (6.67)
  Change at Week 10 | -41.5 (11.05) | -23.3 (23.33)
  Change at Week 11 | -36.9 (12.65) | -26.7 (26.67)
  Change at Week 12 | -38.4 (13.06) | -26.7 (26.67)
  Change at Week 13 | -26.4 (14.24) | -26.7 (26.67)
  Change at Week 14 | -33.7 (13.07) | -26.7 (26.67)
  Change at Week 15 | -41.4 (12.71) | -26.7 (26.67)
  Change at Week 16 | -33.8 (12.37) | -26.7 (26.67)
  Change at Week 17 | -44.0 (11.58) | -26.7 (26.67)
  Change at Week 18 | -51.5 (5.65) | -26.7 (26.67)

11. Secondary Outcome: Change From Baseline in Sleep Loss VAS Over Time
Description: Participants were asked to place a line perpendicular to the VAS line at the point that represents the intensity of their average sleeplessness experienced over the previous 3 nights using a scale from 0 to 10, with 0 indicating no sleeplessness and 10 indicating the worst imaginable sleeplessness at every visit.
Time Frame: Baseline, Weeks 1-8, 10, 12, 14, 16, 18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
units on a scale
  Change at Week 1 | -1.6 (1.12) | 0.1 (0.10) | 0.4 (0.78) | -2.1 (1.17) | -0.4 (0.31) |  | -2.8 (1.81) | 0.1 (NA) — 1 participant in this cohort. | -1.2 (0.25) | -0.1 (0.35)
  Change at Week 2 | -3.1 (1.46) | 0.1 (0.10) | -1.0 (0.60) | -2.6 (0.71) | -0.3 (0.15) |  | -3.4 (1.98) | 0.0 (NA) — 1 participant in this cohort. | -2.1 (0.48) | -0.4 (0.58)
  Change at Week 3 | -2.4 (1.86) | 0.1 (0.10) | -1.6 (0.70) | -3.6 (0.95) | -2.1 (1.49) |  | -4.1 (1.97) | -0.1 (NA) — 1 participant in this cohort. | -3.0 (0.62) | -1.0 (0.75)
  Change at Week 4 | -2.9 (2.30) | 0.1 (0.10) | -1.5 (0.80) | -3.4 (0.86) | -2.9 (1.87) |  | -4.2 (1.81) | -0.1 (NA) — 1 participant in this cohort. | -3.7 (0.62) | -0.3 (1.30)
  Change at Week 5 | -3.5 (2.34) | 0.1 (0.10) | -2.0 (0.72) | -3.9 (0.96) | -3.1 (1.85) |  | -4.4 (1.75) | -2.6 (NA) — 1 participant in this cohort. | -4.0 (0.59) | -1.2 (1.14)
  Change at Week 6 | -2.9 (2.69) | 0.1 (0.10) | -2.3 (0.74) | -3.6 (0.83) | -3.1 (1.85) |  | -5.0 (1.46) | -1.3 (NA) — 1 participant in this cohort. | -4.6 (0.56) | -1.6 (1.20)
  Change at Week 7 | -3.7 (2.16) | 0.0 (0.00) | -2.1 (0.67) | -3.9 (0.79) | -3.4 (1.86) |  | -5.2 (1.33) | -1.0 (NA) — 1 participant in this cohort. | -4.9 (0.58) | -1.8 (1.34)
  Change at Week 8 | -3.3 (2.48) | 0.1 (0.05) | -2.1 (0.67) | -3.8 (0.91) | -3.4 (1.86) |  | -5.3 (1.27) | -1.0 (NA) — 1 participant in this cohort. | -5.4 (0.59) | -2.1 (1.29)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 10 | -3.8 (2.20) | 0.1 (0.10) | -1.7 (0.66) | -5.4 (0.80) | -5.5 (0.90) |  | -5.3 (1.29) | -2.4 (NA) — 1 participant in this cohort. | -5.4 (0.63) | -3.1 (1.36)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -3.3 (2.14) | 0.1 (0.05) | -1.6 (0.73) | -4.3 (0.88) | -5.3 (1.15) |  | -5.2 (1.32) | -2.3 (NA) — 1 participant in this cohort. | -5.2 (0.68) | -3.2 (1.41)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 14 | -3.0 (2.36) | 0.1 (0.10) | -1.7 (0.67) | -4.9 (0.72) | -5.3 (1.15) |  | -5.2 (1.33) | -0.1 (NA) — 1 participant in this cohort. | -5.3 (0.70) | -3.0 (1.49)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -3.5 (2.14) | 0.1 (0.10) | -1.5 (0.78) | -4.0 (1.02) | -5.6 (0.85) |  | -5.4 (1.23) | -0.4 (NA) — 1 participant in this cohort. | -5.1 (0.75) | -2.8 (1.51)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -2.9 (2.28) | 0.1 (0.05) | -1.4 (0.84) | -3.1 (1.03) | -5.7 (2.25) |  | -5.6 (1.11) | -0.6 (NA) — 1 participant in this cohort. | -4.9 (0.90) | -3.3 (1.42)

12. Secondary Outcome: Percent Change From Baseline in Sleep Loss VAS Over Time
Description: as for outcome 11
Time Frame: Baseline, Weeks 1-8, 10, 12, 14, 16, 18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 1: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 1 | -25.1 (20.89) | 2.9 (31.37) | 484.2 (401.19) | 108.2 (483.26) | -5.1 (1.04) |  | -45.5 (27.70) | 22.2 (62.96) | -12.7 (5.20) | -0.3 (7.56)
  Change at Week 2: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 2 | -49.5 (20.04) | 9.9 (30.10) | 12.4 (30.69) | -27.1 (36.97) | -4.1 (2.48) |  | -55.1 (29.83) | 22.1 (67.80) | -23.9 (8.20) | -5.1 (11.91)
  Change at Week 3: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 3 | -38.1 (25.21) | 17.1 (37.85) | 9.9 (44.29) | -47.7 (53.35) | -27.6 (7.82) |  | -66.1 (33.17) | 0.8 (75.41) | -34.7 (7.29) | -16.9 (10.59)
  Change at Week 4: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 4 | -46.8 (28.92) | 22.4 (43.43) | 244.8 (239.53) | 15.4 (288.53) | -38.5 (13.99) |  | -67.0 (28.94) | 4.2 (65.78) | -37.9 (11.30) | 2.4 (16.42)
  Change at Week 5: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 5 | -56.5 (27.85) | 22.2 (41.82) | 8.2 (50.36) | -52.6 (60.66) | -41.1 (17.26) |  | -70.4 (28.63) | -28.9 (65.09) | -47.2 (9.43) | -15.7 (13.70)
  Change at Week 6: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 6 | -47.6 (34.25) | 27.1 (51.43) | -39.8 (14.56) | -61.6 (17.54) | -41.6 (17.91) |  | -79.2 (21.45) | -15.2 (48.76) | -59.4 (8.54) | -21.7 (12.42)
  Change at Week 7: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 7 | -60.0 (22.57) | 19.5 (33.89) | -17.8 (29.08) | -61.5 (35.03) | -45.3 (22.49) |  | -83.1 (18.68) | -14.4 (42.45) | -62.3 (10.19) | -24.3 (14.80)
  Change at Week 8: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 8 | -54.0 (29.23) | 24.2 (43.90) | -26.8 (24.06) | -58.4 (28.98) | -45.3 (22.49) |  | -83.9 (17.07) | -14.3 (38.81) | -69.3 (9.15) | -29.0 (13.29)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 10 | -60.3 (23.36) | 20.9 (35.07) | -43.8 (8.58) | -86.7 (9.51) | -75.0 (0.00) |  | -84.2 (17.92) | -31.1 (40.73) | -68.2 (8.29) | -39.9 (12.85)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -53.6 (13.58) | 23.7 (20.39) | 45.6 (82.52) | -43.2 (91.47) | -71.1 (0.00) |  | -83.4 (18.87) | -30.2 (42.89) | -66.1 (8.84) | -41.9 (13.71)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 14 | -49.5 (19.46) | 27.2 (29.21) | -30.1 (14.43) | -75.6 (15.99) | -71.1 (0.00) |  | -83.0 (19.35) | -6.5 (43.97) | -68.6 (9.28) | -38.0 (14.39)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -57.0 (17.00) | 22.9 (25.53) | -34.4 (15.61) | -69.0 (17.30) | -75.7 (0.00) |  | -85.9 (16.02) | -8.9 (36.40) | -66.0 (9.77) | -36.7 (15.16)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -47.3 (11.94) | 27.7 (17.93) | -23.3 (15.15) | -56.1 (16.79) | -74.7 (0.00) |  | -89.9 (11.26) | -9.8 (25.59) | -61.6 (11.11) | -43.6 (17.22)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 1; Test type: Superiority; p = 0.5403, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.9, 80% CI 2-sided [-94.32 to 38.46], Standard Error of Mean 40.54
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 1; Test type: Superiority; p = 0.5587, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 376.1, 80% CI 2-sided [-462.83 to 1214.97], Standard Error of Mean 631.83
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 1; Test type: Superiority; p = 0.4516, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -67.7, 80% CI 2-sided [-205.33 to 69.93], Standard Error of Mean 72.99
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 1; Test type: Superiority; p = 0.2052, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -12.5, 80% CI 2-sided [-25.13 to 0.15], Standard Error of Mean 9.50
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 2; Test type: Superiority; p = 0.2240, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -59.4, 80% CI 2-sided [-123.09 to 4.28], Standard Error of Mean 38.89
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 2; Test type: Superiority; p = 0.4242, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 39.5, 80% CI 2-sided [-24.70 to 103.65], Standard Error of Mean 48.33
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 2; Test type: Superiority; p = 0.4295, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -77.2, 80% CI 2-sided [-225.44 to 71.01], Standard Error of Mean 78.61
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 2; Test type: Superiority; p = 0.2272, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -18.7, 80% CI 2-sided [-38.64 to 1.20], Standard Error of Mean 14.97
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 3; Test type: Superiority; p = 0.3416, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -55.1, 80% CI 2-sided [-135.23 to 24.95], Standard Error of Mean 48.90
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 3; Test type: Superiority; p = 0.4192, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 57.6, 80% CI 2-sided [-35.02 to 150.19], Standard Error of Mean 69.75
Statistical Analysis 11: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 3; Test type: Superiority; p = 0.5245, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -66.8, 80% CI 2-sided [-231.66 to 98.02], Standard Error of Mean 87.42
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 3; Test type: Superiority; p = 0.1988, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -17.8, 80% CI 2-sided [-35.47 to -0.05], Standard Error of Mean 13.31
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.3054, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -69.2, 80% CI 2-sided [-161.08 to 22.72], Standard Error of Mean 56.11
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.5504, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 229.4, 80% CI 2-sided [-271.51 to 730.22], Standard Error of Mean 377.23
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.4493, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -71.2, 80% CI 2-sided [-214.96 to 72.65], Standard Error of Mean 76.27
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0665, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -40.3, 80% CI 2-sided [-67.74 to -12.85], Standard Error of Mean 20.63
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 5; Test type: Superiority; p = 0.2411, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -78.7, 80% CI 2-sided [-167.25 to 9.75], Standard Error of Mean 54.04
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 5; Test type: Superiority; p = 0.4528, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 60.8, 80% CI 2-sided [-44.51 to 166.08], Standard Error of Mean 79.30
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 5; Test type: Superiority; p = 0.6381, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -41.4, 80% CI 2-sided [-183.72 to 100.85], Standard Error of Mean 75.46
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 5; Test type: Superiority; p = 0.0837, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -31.5, 80% CI 2-sided [-54.44 to -8.62], Standard Error of Mean 17.22
Statistical Analysis 21: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 6; Test type: Superiority; p = 0.3428, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -74.7, 80% CI 2-sided [-183.53 to 34.13], Standard Error of Mean 66.45
Statistical Analysis 22: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 6; Test type: Superiority; p = 0.3533, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 21.8, 80% CI 2-sided [-8.63 to 52.27], Standard Error of Mean 22.93
Statistical Analysis 23: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 6; Test type: Superiority; p = 0.3755, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -63.9, 80% CI 2-sided [-170.51 to 42.66], Standard Error of Mean 56.53
Statistical Analysis 24: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 6; Test type: Superiority; p = 0.0268, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -37.6, 80% CI 2-sided [-58.39 to -16.87], Standard Error of Mean 15.60
Statistical Analysis 25: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 7; Test type: Superiority; p = 0.1672, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -79.5, 80% CI 2-sided [-151.20 to -7.75], Standard Error of Mean 43.79
Statistical Analysis 26: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 7; Test type: Superiority; p = 0.3518, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 43.7, 80% CI 2-sided [-17.09 to 104.55], Standard Error of Mean 45.81
Statistical Analysis 27: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 7; Test type: Superiority; p = 0.2974, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -68.7, 80% CI 2-sided [-161.52 to 24.09], Standard Error of Mean 49.22
Statistical Analysis 28: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 7; Test type: Superiority; p = 0.0555, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -38.1, 80% CI 2-sided [-62.83 to -13.33], Standard Error of Mean 18.60
Statistical Analysis 29: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.2614, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -78.3, 80% CI 2-sided [-171.17 to 14.62], Standard Error of Mean 56.72
Statistical Analysis 30: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.4134, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 31.7, 80% CI 2-sided [-18.62 to 81.98], Standard Error of Mean 37.89
Statistical Analysis 31: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.2620, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -69.6, 80% CI 2-sided [-154.44 to 15.24], Standard Error of Mean 44.99
Statistical Analysis 32: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0269, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -40.2, 80% CI 2-sided [-62.46 to -18.02], Standard Error of Mean 16.70
Statistical Analysis 33: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 10; Test type: Superiority; p = 0.1709, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -81.2, 80% CI 2-sided [-155.46 to -7.02], Standard Error of Mean 45.32
Statistical Analysis 34: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 10; Test type: Superiority; p = 0.0042, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 42.9, 80% CI 2-sided [25.61 to 60.22], Standard Error of Mean 12.98
Statistical Analysis 35: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 10; Test type: Superiority; p = 0.3772, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -53.2, 80% CI 2-sided [-142.19 to 35.88], Standard Error of Mean 47.22
Statistical Analysis 36: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 10; Test type: Superiority; p = 0.0857, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -28.3, 80% CI 2-sided [-49.06 to -7.63], Standard Error of Mean 15.54
Statistical Analysis 37: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.0607, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -77.3, 80% CI 2-sided [-120.48 to -34.20], Standard Error of Mean 26.34
Statistical Analysis 38: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.4862, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 88.8, 80% CI 2-sided [-77.57 to 255.22], Standard Error of Mean 124.79
Statistical Analysis 39: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 12; Test type: Superiority; p = 0.3968, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -53.2, 80% CI 2-sided [-146.96 to 40.58], Standard Error of Mean 49.73
Statistical Analysis 40: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.1624, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -24.2, 80% CI 2-sided [-46.31 to -2.11], Standard Error of Mean 16.57
Statistical Analysis 41: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 14; Test type: Superiority; p = 0.1349, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -76.8, 80% CI 2-sided [-138.58 to -14.93], Standard Error of Mean 37.75
Statistical Analysis 42: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 14; Test type: Superiority; p = 0.0525, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 45.5, 80% CI 2-sided [16.38 to 74.56], Standard Error of Mean 21.81
Statistical Analysis 43: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 14; Test type: Superiority; p = 0.2719, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -76.6, 80% CI 2-sided [-172.71 to 19.55], Standard Error of Mean 50.98
Statistical Analysis 44: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 14; Test type: Superiority; p = 0.0957, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -30.7, 80% CI 2-sided [-53.86 to -7.49], Standard Error of Mean 17.39
Statistical Analysis 45: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.0942, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -79.8, 80% CI 2-sided [-133.83 to -25.78], Standard Error of Mean 32.98
Statistical Analysis 46: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.1606, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 34.6, 80% CI 2-sided [3.16 to 66.09], Standard Error of Mean 23.60
Statistical Analysis 47: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.2096, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -77.0, 80% CI 2-sided [-156.58 to 2.58], Standard Error of Mean 42.20
Statistical Analysis 48: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.1279, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -29.3, 80% CI 2-sided [-53.74 to -4.89], Standard Error of Mean 18.32
Statistical Analysis 49: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.0479, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -75.0, 80% CI 2-sided [-112.96 to -37.08], Standard Error of Mean 23.17
Statistical Analysis 50: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Superiority; p = 0.1700, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 32.8, 80% CI 2-sided [2.28 to 63.37], Standard Error of Mean 22.91
Statistical Analysis 51: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.1142, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -80.1, 80% CI 2-sided [-136.03 to -24.15], Standard Error of Mean 29.67
Statistical Analysis 52: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Superiority; p = 0.3980, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -18.0, 80% CI 2-sided [-45.80 to 9.71], Standard Error of Mean 20.82

13. Secondary Outcome: Change From Baseline in Weekly Average of Difficulty Falling Asleep Numerical Rating Scale (NRS) Over Time
Description: Participants were asked daily to assign a numerical score to the intensity of their difficulty falling asleep last night due to itch using a scale from 0 to 10, with 0 indicating not difficult at all and 10 indicating extremely difficult.
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
score on a scale
  Change at Week 1 | -2.1 (0.67) | -0.3 (0.29) | -0.6 (0.44) | -1.7 (0.40) | -0.3 (0.08) |  | -3.0 (1.31) | -1.0 (NA) — 1 participant in this cohort. | -0.7 (0.16) | 0.0 (0.24)
  Change at Week 2 | -3.3 (0.78) | -0.4 (0.43) | -2.0 (0.52) | -3.1 (0.57) | -0.9 (0.30) |  | -4.3 (1.96) | -1.0 (NA) — 1 participant in this cohort. | -1.3 (0.26) | -0.6 (0.35)
  Change at Week 3 | -4.2 (1.21) | -0.5 (0.50) | -2.6 (0.59) | -2.9 (0.70) | -1.6 (0.87) |  | -4.6 (2.10) | -1.6 (NA) — 1 participant in this cohort. | -2.4 (0.56) | -0.8 (0.42)
  Change at Week 4 | -4.5 (1.35) | 0.0 (0.00) | -2.7 (0.72) | -2.9 (0.82) | -2.5 (1.57) |  | -4.8 (1.91) | -2.1 (NA) — 1 participant in this cohort. | -3.1 (0.55) | -1.0 (0.70)
  Change at Week 5 | -5.0 (1.57) | -0.4 (0.43) | -3.0 (0.76) | -3.0 (0.71) | -2.9 (1.64) |  | -5.2 (1.95) | -2.0 (NA) — 1 participant in this cohort. | -4.1 (0.72) | -1.5 (0.89)
  Change at Week 6 | -5.0 (1.45) | -0.5 (0.50) | -3.0 (0.69) | -3.8 (0.71) | -3.1 (1.61) |  | -5.5 (1.82) | -2.6 (NA) — 1 participant in this cohort. | -4.4 (0.69) | -1.4 (0.90)
  Change at Week 7 | -4.5 (1.56) | -0.2 (0.21) | -3.0 (0.65) | -3.7 (0.75) | -3.6 (1.65) |  | -5.6 (1.76) | -2.6 (NA) — 1 participant in this cohort. | -4.8 (0.72) | -1.8 (1.08)
  Change at Week 8 | -3.8 (1.66) | -0.3 (0.29) | -3.2 (0.64) | -2.9 (0.81) | -3.6 (1.65) |  | -5.4 (1.94) | -3.3 (NA) — 1 participant in this cohort. | -5.2 (0.70) | -2.1 (1.21)
  Change at Week 9: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 9 | -4.4 (1.46) | 0.7 (0.71) | -2.9 (0.69) | -3.7 (0.65) | -5.1 (0.86) |  | -5.4 (1.88) | -3.4 (NA) — 1 participant in this cohort. | -5.3 (0.70) | -2.4 (1.27)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 10 | -4.4 (1.64) | -0.5 (0.50) | -2.6 (0.65) | -4.5 (0.55) | -5.1 (0.86) |  | -5.6 (1.69) | -3.0 (NA) — 1 participant in this cohort. | -5.2 (0.77) | -2.4 (1.21)
  Change at Week 11: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 11 | -4.7 (1.78) | -0.5 (0.50) | -2.6 (0.76) | -4.6 (0.69) | -5.1 (0.86) |  | -5.7 (1.61) | -3.1 (NA) — 1 participant in this cohort. | -5.0 (0.77) | -2.4 (1.20)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 12 | -4.7 (1.73) | -0.5 (0.50) | -2.5 (0.73) | -4.1 (0.71) | -5.1 (0.86) |  | -5.9 (1.50) | -2.6 (NA) — 1 participant in this cohort. | -4.9 (0.78) | -2.5 (1.17)
  Change at Week 13: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 13 | -4.1 (1.90) | -0.5 (0.50) | -2.5 (0.65) | -4.3 (0.73) | -5.6 (0.43) |  | -5.9 (1.53) | -1.9 (NA) — 1 participant in this cohort. | -5.0 (0.80) | -2.5 (1.18)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 14 | -3.6 (1.92) | -0.5 (0.50) | -2.8 (0.65) | -4.3 (0.78) | -5.6 (0.36) |  | -5.8 (1.58) | -2.1 (NA) — 1 participant in this cohort. | -5.1 (0.78) | -2.6 (1.20)
  Change at Week 15: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 15 | -4.4 (1.77) | -0.5 (0.50) | -2.6 (0.61) | -4.1 (0.73) | -5.6 (0.36) |  | -6.0 (1.45) | -2.4 (NA) — 1 participant in this cohort. | -5.0 (0.83) | -2.8 (1.35)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 16 | -4.1 (1.86) | -0.5 (0.50) | -2.8 (0.68) | -3.8 (0.91) | -5.6 (0.36) |  | -6.0 (1.43) | -1.9 (NA) — 1 participant in this cohort. | -4.9 (0.81) | -2.7 (1.32)
  Change at Week 17: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 17 | -4.2 (1.91) | -0.5 (0.50) | -2.7 (0.64) | -3.5 (0.85) | -5.6 (0.36) |  | -6.2 (1.32) | -1.4 (NA) — 1 participant in this cohort. | -4.6 (0.97) | -3.0 (1.37)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 18 | -4.4 (1.79) | -0.5 (0.50) | -2.8 (0.72) | -3.6 (0.92) | -5.7 (0.43) |  | -6.2 (1.32) | -1.3 (NA) — 1 participant in this cohort. | -4.6 (0.98) | -3.0 (1.36)

14. Secondary Outcome: Percent Change From Baseline in Weekly Average of Difficulty Falling Asleep NRS Over Time
Description: as for outcome 13
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 1: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 1 | -35.3 (9.68) | -22.2 (13.83) | -4.9 (8.21) | -26.6 (9.88) | -3.6 (1.17) |  | -42.9 (17.69) | -7.4 (36.83) | -9.3 (2.32) | 1.2 (3.33)
  Change at Week 2: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 2 | -51.1 (13.32) | -34.9 (19.03) | -31.2 (7.80) | -48.7 (9.38) | -10.9 (5.13) |  | -59.3 (23.10) | -0.5 (48.09) | -15.0 (3.50) | -9.3 (5.03)
  Change at Week 3: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 3 | -63.9 (20.16) | -40.9 (28.80) | -42.1 (8.81) | -48.7 (10.60) | -20.0 (15.28) |  | -64.8 (24.87) | -6.2 (51.77) | -27.6 (6.38) | -11.2 (9.16)
  Change at Week 4: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 4 | -61.0 (15.91) | -1.4 (22.72) | -43.3 (10.71) | -50.3 (12.88) | -31.4 (27.58) |  | -67.6 (21.14) | -14.2 (44.00) | -36.3 (6.64) | -12.2 (9.53)
  Change at Week 5: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 5 | -71.7 (22.82) | -36.4 (32.59) | -46.0 (11.47) | -50.4 (13.80) | -37.2 (28.02) |  | -73.1 (23.65) | -15.4 (49.24) | -48.4 (7.51) | -20.8 (10.78)
  Change at Week 6: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 6 | -73.1 (21.37) | -42.1 (30.52) | -47.5 (9.49) | -60.6 (11.42) | -39.8 (26.65) |  | -79.0 (25.98) | -30.3 (54.08) | -52.7 (7.40) | -19.0 (10.63)
  Change at Week 7: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 7 | -62.2 (19.51) | -19.4 (27.88) | -50.5 (8.27) | -61.5 (9.95) | -46.3 (23.22) |  | -80.0 (24.71) | -30.3 (51.45) | -57.2 (8.21) | -24.5 (11.79)
  Change at Week 8: number analyzed (Participants) | 4 | 2 | 13 | 9 | 3 | 0 | 4 | 1 | 14 | 7
  Change at Week 8 | -51.9 (21.00) | -25.8 (30.00) | -54.1 (8.75) | -47.9 (10.52) | -46.3 (23.22) |  | -77.0 (28.52) | -38.6 (59.36) | -63.2 (8.55) | -27.5 (12.29)
  Change at Week 9: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 9 | -52.4 (10.60) | 55.9 (15.15) | -50.6 (8.32) | -60.6 (9.20) | -66.9 (0.00) |  | -78.0 (27.25) | -40.3 (56.72) | -64.3 (8.48) | -32.3 (12.17)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 10 | -62.3 (22.58) | -43.1 (32.26) | -45.5 (7.86) | -69.4 (8.70) | -66.9 (0.00) |  | -80.6 (23.28) | -35.5 (48.46) | -62.0 (8.70) | -31.5 (12.50)
  Change at Week 11: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 11 | -66.4 (24.89) | -43.1 (35.55) | -43.2 (9.82) | -69.8 (10.86) | -66.9 (0.00) |  | -82.1 (21.38) | -37.1 (44.50) | -58.9 (8.47) | -33.2 (12.17)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 12 | -66.4 (23.94) | -43.1 (34.20) | -43.4 (10.02) | -64.0 (11.08) | -66.9 (0.00) |  | -85.2 (18.38) | -30.2 (38.26) | -58.5 (8.78) | -33.7 (12.60)
  Change at Week 13: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 13 | -55.7 (26.31) | -43.7 (37.59) | -43.5 (9.52) | -68.2 (10.53) | -72.8 (0.00) |  | -84.6 (19.01) | -21.9 (39.57) | -60.6 (9.18) | -34.1 (13.19)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 14 | -48.5 (25.78) | -44.0 (36.83) | -49.4 (9.01) | -68.9 (9.97) | -73.8 (0.00) |  | -83.6 (20.28) | -25.2 (42.21) | -61.7 (9.25) | -34.1 (13.28)
  Change at Week 15: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 15 | -62.3 (24.47) | -43.3 (34.96) | -44.1 (8.74) | -67.0 (9.67) | -73.8 (0.00) |  | -86.2 (17.11) | -28.5 (35.62) | -60.2 (9.90) | -38.3 (14.22)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 16 | -56.4 (25.57) | -43.7 (36.52) | -47.8 (10.02) | -64.3 (11.08) | -73.8 (0.00) |  | -86.7 (16.48) | -21.8 (34.30) | -58.9 (9.71) | -37.0 (13.95)
  Change at Week 17: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 17 | -58.5 (26.89) | -43.6 (38.41) | -45.1 (9.46) | -60.3 (10.47) | -73.8 (0.00) |  | -89.3 (13.31) | -16.8 (27.70) | -53.7 (11.52) | -41.2 (16.54)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 11 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 18 | -61.1 (24.70) | -43.4 (35.29) | -48.1 (10.22) | -61.9 (11.30) | -74.7 (0.00) |  | -89.3 (13.31) | -15.1 (27.70) | -53.4 (11.61) | -41.8 (16.68)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 1; Test type: Superiority; p = 0.4979, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -13.2, 80% CI 2-sided [-41.17 to 14.86], Standard Error of Mean 17.11
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 1; Test type: Superiority; p = 0.1079, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 21.7, 80% CI 2-sided [4.63 to 38.83], Standard Error of Mean 12.88
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 1; Test type: Superiority; p = 0.4837, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -35.6, 80% CI 2-sided [-114.19 to 43.07], Standard Error of Mean 41.70
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 1; Test type: Superiority; p = 0.0208, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -10.5, 80% CI 2-sided [-15.99 to -4.98], Standard Error of Mean 4.14
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 2; Test type: Superiority; p = 0.5413, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -16.2, 80% CI 2-sided [-54.74 to 22.38], Standard Error of Mean 23.54
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 2; Test type: Superiority; p = 0.1683, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 17.5, 80% CI 2-sided [1.28 to 33.74], Standard Error of Mean 12.22
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 2; Test type: Superiority; p = 0.3933, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -58.8, 80% CI 2-sided [-161.43 to 43.89], Standard Error of Mean 54.45
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 2; Test type: Superiority; p = 0.3705, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -5.7, 80% CI 2-sided [-14.06 to 2.58], Standard Error of Mean 6.25
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 3; Test type: Superiority; p = 0.5644, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -23.0, 80% CI 2-sided [-81.36 to 35.34], Standard Error of Mean 35.63
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 3; Test type: Superiority; p = 0.6384, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 6.6, 80% CI 2-sided [-11.75 to 24.94], Standard Error of Mean 13.82
Statistical Analysis 11: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 3; Test type: Superiority; p = 0.4229, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -58.6, 80% CI 2-sided [-169.13 to 51.95], Standard Error of Mean 58.62
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 3; Test type: Superiority; p = 0.1688, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -16.3, 80% CI 2-sided [-31.47 to -1.18], Standard Error of Mean 11.38
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.1243, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -59.6, 80% CI 2-sided [-105.59 to -13.53], Standard Error of Mean 28.11
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.6841, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 6.9, 80% CI 2-sided [-15.35 to 29.22], Standard Error of Mean 16.79
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.3963, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -53.4, 80% CI 2-sided [-147.31 to 40.59], Standard Error of Mean 49.83
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0571, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -24.1, 80% CI 2-sided [-39.85 to -8.32], Standard Error of Mean 11.85
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 5; Test type: Superiority; p = 0.4457, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -35.3, 80% CI 2-sided [-101.32 to 30.73], Standard Error of Mean 40.32
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 5; Test type: Superiority; p = 0.8075, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 4.4, 80% CI 2-sided [-19.44 to 28.32], Standard Error of Mean 17.99
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 5; Test type: Superiority; p = 0.4093, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -57.7, 80% CI 2-sided [-162.84 to 47.40], Standard Error of Mean 55.75
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 5; Test type: Superiority; p = 0.0543, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.6, 80% CI 2-sided [-45.42 to -9.76], Standard Error of Mean 13.40
Statistical Analysis 21: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 6; Test type: Superiority; p = 0.4711, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -31.0, 80% CI 2-sided [-92.88 to 30.78], Standard Error of Mean 37.75
Statistical Analysis 22: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 6; Test type: Superiority; p = 0.3925, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 13.0, 80% CI 2-sided [-6.74 to 32.79], Standard Error of Mean 14.89
Statistical Analysis 23: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 6; Test type: Superiority; p = 0.5095, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -48.7, 80% CI 2-sided [-164.22 to 66.72], Standard Error of Mean 61.24
Statistical Analysis 24: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 6; Test type: Superiority; p = 0.0199, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -33.8, 80% CI 2-sided [-51.35 to -16.18], Standard Error of Mean 13.22
Statistical Analysis 25: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 7; Test type: Superiority; p = 0.3029, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -42.8, 80% CI 2-sided [-99.26 to 13.69], Standard Error of Mean 34.48
Statistical Analysis 26: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 7; Test type: Superiority; p = 0.4094, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 10.9, 80% CI 2-sided [-6.28 to 28.16], Standard Error of Mean 12.97
Statistical Analysis 27: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 7; Test type: Superiority; p = 0.4828, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -49.8, 80% CI 2-sided [-159.63 to 60.05], Standard Error of Mean 58.25
Statistical Analysis 28: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 7; Test type: Superiority; p = 0.0383, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -32.8, 80% CI 2-sided [-52.26 to -13.26], Standard Error of Mean 14.66
Statistical Analysis 29: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.5322, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -26.1, 80% CI 2-sided [-86.66 to 34.65], Standard Error of Mean 37.10
Statistical Analysis 30: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.6577, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -6.2, 80% CI 2-sided [-24.38 to 12.03], Standard Error of Mean 13.71
Statistical Analysis 31: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.6259, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -38.3, 80% CI 2-sided [-165.08 to 88.40], Standard Error of Mean 67.21
Statistical Analysis 32: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0312, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -35.7, 80% CI 2-sided [-56.01 to -15.38], Standard Error of Mean 15.27
Statistical Analysis 33: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 9; Test type: Superiority; p = 0.0103, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -108.3, 80% CI 2-sided [-138.97 to -77.61], Standard Error of Mean 18.73
Statistical Analysis 34: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 9; Test type: Superiority; p = 0.4330, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 10.0, 80% CI 2-sided [-6.59 to 26.56], Standard Error of Mean 12.43
Statistical Analysis 35: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 9; Test type: Superiority; p = 0.6165, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -37.7, 80% CI 2-sided [-158.82 to 83.39], Standard Error of Mean 64.23
Statistical Analysis 36: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 9; Test type: Superiority; p = 0.0488, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -32.0, 80% CI 2-sided [-52.11 to -11.84], Standard Error of Mean 15.13
Statistical Analysis 37: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 10; Test type: Superiority; p = 0.6636, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -19.2, 80% CI 2-sided [-84.53 to 46.16], Standard Error of Mean 39.90
Statistical Analysis 38: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 10; Test type: Superiority; p = 0.0583, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 23.9, 80% CI 2-sided [8.18 to 39.52], Standard Error of Mean 11.75
Statistical Analysis 39: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 10; Test type: Superiority; p = 0.4975, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -45.1, 80% CI 2-sided [-148.55 to 58.36], Standard Error of Mean 54.87
Statistical Analysis 40: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 10; Test type: Superiority; p = 0.0653, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -30.5, 80% CI 2-sided [-51.17 to -9.82], Standard Error of Mean 15.54
Statistical Analysis 41: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 11; Test type: Superiority; p = 0.6316, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -23.4, 80% CI 2-sided [-95.42 to 48.62], Standard Error of Mean 43.98
Statistical Analysis 42: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 11; Test type: Superiority; p = 0.0874, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 26.6, 80% CI 2-sided [7.05 to 46.18], Standard Error of Mean 14.68
Statistical Analysis 43: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 11; Test type: Superiority; p = 0.4662, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -45.0, 80% CI 2-sided [-139.99 to 50.03], Standard Error of Mean 50.39
Statistical Analysis 44: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 11; Test type: Superiority; p = 0.1073, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -25.6, 80% CI 2-sided [-45.76 to -5.51], Standard Error of Mean 15.12
Statistical Analysis 45: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.6197, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -23.3, 80% CI 2-sided [-92.62 to 45.96], Standard Error of Mean 42.31
Statistical Analysis 46: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.1868, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 20.6, 80% CI 2-sided [0.63 to 40.55], Standard Error of Mean 14.97
Statistical Analysis 47: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 12; Test type: Superiority; p = 0.3321, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -55.0, 80% CI 2-sided [-136.65 to 26.71], Standard Error of Mean 43.32
Statistical Analysis 48: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.1310, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -24.8, 80% CI 2-sided [-45.64 to -3.95], Standard Error of Mean 15.67
Statistical Analysis 49: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 13; Test type: Superiority; p = 0.8128, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -12.0, 80% CI 2-sided [-88.15 to 64.13], Standard Error of Mean 46.49
Statistical Analysis 50: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 13; Test type: Superiority; p = 0.1004, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 24.7, 80% CI 2-sided [5.75 to 43.69], Standard Error of Mean 14.23
Statistical Analysis 51: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 13; Test type: Superiority; p = 0.2962, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -62.8, 80% CI 2-sided [-147.28 to 21.71], Standard Error of Mean 44.81
Statistical Analysis 52: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 13; Test type: Superiority; p = 0.1236, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -26.5, 80% CI 2-sided [-48.31 to -4.67], Standard Error of Mean 16.40
Statistical Analysis 53: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 14; Test type: Superiority; p = 0.9276, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -4.5, 80% CI 2-sided [-79.10 to 70.11], Standard Error of Mean 45.55
Statistical Analysis 54: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 14; Test type: Superiority; p = 0.1657, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 19.5, 80% CI 2-sided [1.55 to 37.45], Standard Error of Mean 13.46
Statistical Analysis 55: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 14; Test type: Superiority; p = 0.3461, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -58.4, 80% CI 2-sided [-148.54 to 31.71], Standard Error of Mean 47.80
Statistical Analysis 56: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 14; Test type: Superiority; p = 0.1118, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.6, 80% CI 2-sided [-49.58 to -5.64], Standard Error of Mean 16.51
Statistical Analysis 57: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 15; Test type: Superiority; p = 0.6912, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -18.9, 80% CI 2-sided [-89.75 to 51.89], Standard Error of Mean 43.24
Statistical Analysis 58: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 15; Test type: Superiority; p = 0.0973, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 22.9, 80% CI 2-sided [5.50 to 40.35], Standard Error of Mean 13.07
Statistical Analysis 59: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 15; Test type: Superiority; p = 0.2890, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -57.7, 80% CI 2-sided [-133.72 to 18.37], Standard Error of Mean 40.33
Statistical Analysis 60: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 15; Test type: Superiority; p = 0.2310, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -21.9, 80% CI 2-sided [-45.43 to 1.60], Standard Error of Mean 17.68
Statistical Analysis 61: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.7967, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -12.7, 80% CI 2-sided [-86.69 to 61.28], Standard Error of Mean 45.17
Statistical Analysis 62: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.2868, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 16.5, 80% CI 2-sided [-3.50 to 36.44], Standard Error of Mean 14.98
Statistical Analysis 63: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.2369, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -64.9, 80% CI 2-sided [-138.08 to 8.37], Standard Error of Mean 38.83
Statistical Analysis 64: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.2228, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -21.9, 80% CI 2-sided [-44.97 to 1.17], Standard Error of Mean 17.34
Statistical Analysis 65: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 17; Test type: Superiority; p = 0.7740, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -14.9, 80% CI 2-sided [-92.74 to 62.89], Standard Error of Mean 47.51
Statistical Analysis 66: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 17; Test type: Superiority; p = 0.3000, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 15.1, 80% CI 2-sided [-3.74 to 33.98], Standard Error of Mean 14.14
Statistical Analysis 67: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 17; Test type: Superiority; p = 0.1472, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -72.4, 80% CI 2-sided [-131.59 to -13.30], Standard Error of Mean 31.37
Statistical Analysis 68: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 17; Test type: Superiority; p = 0.5536, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -12.4, 80% CI 2-sided [-39.77 to 14.94], Standard Error of Mean 20.56
Statistical Analysis 69: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.7131, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -17.6, 80% CI 2-sided [-89.13 to 53.84], Standard Error of Mean 43.65
Statistical Analysis 70: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Superiority; p = 0.3762, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 13.9, 80% CI 2-sided [-6.49 to 34.24], Standard Error of Mean 15.27
Statistical Analysis 71: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.1419, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -74.1, 80% CI 2-sided [-133.26 to -14.97], Standard Error of Mean 31.37
Statistical Analysis 72: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Superiority; p = 0.5817, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -11.6, 80% CI 2-sided [-39.22 to 15.95], Standard Error of Mean 20.74

15. Secondary Outcome: Change From Baseline in Weekly Average of Sleep Quality NRS Over Time
Description: Participants were asked daily to assign a numerical score to the quality of their sleep in the previous night using a scale from 0 to 10, with 0 indicating best possible sleep and 10 indicating worst possible sleep.
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
score on a scale
  Change at Week 1 | -0.8 (1.32) | -0.3 (0.29) | -0.2 (0.33) | -1.6 (0.43) | -0.2 (0.17) |  | -2.6 (1.26) | -1.0 (NA) — 1 participant in this cohort. | -0.6 (0.20) | -0.3 (0.19)
  Change at Week 2 | -2.0 (1.63) | -0.4 (0.43) | -1.7 (0.56) | -2.7 (0.60) | -0.7 (0.41) |  | -3.7 (1.75) | -0.7 (NA) — 1 participant in this cohort. | -1.1 (0.30) | -0.4 (0.29)
  Change at Week 3 | -1.9 (1.86) | -0.5 (0.50) | -1.9 (0.54) | -2.7 (0.62) | -1.5 (1.02) |  | -4.2 (1.98) | -1.0 (NA) — 1 participant in this cohort. | -2.0 (0.52) | -0.5 (0.42)
  Change at Week 4 | -2.6 (2.12) | 0.0 (0.00) | -2.0 (0.65) | -2.7 (0.93) | -2.3 (1.67) |  | -4.4 (1.78) | -2.0 (NA) — 1 participant in this cohort. | -2.8 (0.59) | -0.9 (0.64)
  Change at Week 5 | -2.8 (2.35) | -0.4 (0.43) | -2.3 (0.68) | -2.8 (0.73) | -2.8 (1.75) |  | -4.4 (1.61) | -1.9 (NA) — 1 participant in this cohort. | -3.5 (0.75) | -1.2 (0.91)
  Change at Week 6 | -2.6 (2.45) | -0.5 (0.50) | -2.4 (0.69) | -3.7 (0.64) | -3.0 (1.73) |  | -5.2 (1.53) | -2.4 (NA) — 1 participant in this cohort. | -3.8 (0.70) | -1.1 (0.95)
  Change at Week 7 | -2.6 (2.31) | -0.2 (0.21) | -2.4 (0.65) | -3.6 (0.79) | -3.4 (1.78) |  | -5.3 (1.43) | -2.0 (NA) — 1 participant in this cohort. | -4.2 (0.71) | -1.5 (1.10)
  Change at Week 8 | -2.5 (2.38) | -0.3 (0.29) | -2.5 (0.67) | -3.6 (0.89) | -3.4 (1.78) |  | -5.6 (1.24) | -3.0 (NA) — 1 participant in this cohort. | -4.7 (0.72) | -1.8 (1.23)
  Change at Week 9: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 9 | -2.9 (2.12) | 0.7 (0.71) | -2.3 (0.69) | -4.1 (0.78) | -5.1 (0.86) |  | -5.6 (1.28) | -3.0 (NA) — 1 participant in this cohort. | -5.0 (0.70) | -2.0 (1.35)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 10 | -2.5 (2.23) | -0.5 (0.50) | -1.9 (0.65) | -4.9 (0.71) | -5.1 (0.86) |  | -5.7 (1.21) | -2.6 (NA) — 1 participant in this cohort. | -5.2 (0.74) | -1.9 (1.29)
  Change at Week 11: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 11 | -2.5 (1.93) | -0.5 (0.50) | -2.0 (0.72) | -4.9 (0.77) | -5.1 (0.86) |  | -5.7 (1.21) | -2.9 (NA) — 1 participant in this cohort. | -4.9 (0.78) | -2.0 (1.25)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 12 | -2.7 (2.04) | -0.5 (0.50) | -1.6 (0.80) | -4.4 (0.83) | -5.1 (0.86) |  | -5.7 (1.21) | -2.7 (NA) — 1 participant in this cohort. | -4.8 (0.80) | -2.0 (1.24)
  Change at Week 13: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 13 | -2.4 (2.11) | -0.5 (0.50) | -1.9 (0.72) | -4.6 (0.85) | -5.6 (0.43) |  | -5.6 (1.24) | -1.7 (NA) — 1 participant in this cohort. | -5.0 (0.80) | -2.1 (1.24)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 14 | -2.5 (2.43) | -0.5 (0.50) | -2.0 (0.62) | -4.3 (0.94) | -5.6 (0.36) |  | -5.5 (1.30) | -1.9 (NA) — 1 participant in this cohort. | -5.0 (0.77) | -5.0 (0.81)
  Change at Week 15: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 15 | -2.6 (2.31) | -0.5 (0.50) | -2.1 (0.62) | -4.1 (0.89) | -5.6 (0.36) |  | -5.7 (1.22) | -2.1 (NA) — 1 participant in this cohort. | -5.0 (0.81) | -2.3 (1.27)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 16 | -3.0 (2.23) | -0.5 (0.50) | -2.5 (0.70) | -3.6 (1.01) | -5.6 (0.36) |  | -5.8 (1.19) | -1.4 (NA) — 1 participant in this cohort. | -4.9 (0.80) | -2.2 (1.25)
  Change at Week 17: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 17 | -3.5 (2.03) | -0.5 (0.50) | -2.3 (0.66) | -3.7 (0.98) | -5.6 (0.36) |  | -5.7 (1.21) | -1.4 (NA) — 1 participant in this cohort. | -4.6 (0.95) | -2.5 (1.29)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 18 | -3.3 (2.12) | -0.5 (0.50) | -2.3 (0.74) | -3.6 (1.00) | -5.7 (0.43) |  | -5.7 (1.21) | -1.3 (NA) — 1 participant in this cohort. | -4.6 (0.96) | -2.5 (1.29)

16. Secondary Outcome: Percent Change From Baseline in Weekly Average of Sleep Quality NRS Over Time
Description: as for outcome 15
Time Frame: Baseline, Weeks 1-18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 1 | -1.0 (32.15) | -28.7 (45.50) | -2.6 (5.75) | -26.3 (7.18) | -3.0 (2.92) |  | -40.7 (17.63) | -1.4 (38.74) | -6.7 (2.75) | -4.9 (3.91)
  Change at Week 2 | -20.2 (34.79) | -42.6 (49.24) | -28.7 (8.26) | -45.6 (10.32) | -9.2 (7.29) |  | -56.7 (24.07) | 6.8 (52.89) | -12.4 (3.67) | -6.0 (5.22)
  Change at Week 3 | -15.5 (39.26) | -49.7 (55.57) | -33.4 (7.94) | -47.2 (9.92) | -18.9 (17.50) |  | -64.4 (26.92) | 6.3 (59.14) | -22.7 (6.03) | -7.1 (8.58)
  Change at Week 4 | -25.0 (31.15) | -2.2 (44.09) | -34.6 (10.18) | -47.9 (12.72) | -29.8 (28.43) |  | -67.2 (22.95) | -6.6 (50.42) | -34.4 (6.75) | -11.7 (9.60)
  Change at Week 5 | -25.7 (42.76) | -43.4 (60.51) | -38.4 (9.11) | -50.7 (11.38) | -35.5 (30.62) |  | -67.3 (23.31) | -16.9 (51.21) | -43.0 (7.95) | -15.9 (11.31)
  Change at Week 6 | -20.9 (47.36) | -50.4 (67.03) | -40.9 (8.43) | -62.7 (10.54) | -38.1 (30.62) |  | -80.2 (22.99) | -32.7 (50.51) | -46.7 (7.82) | -13.0 (11.12)
  Change at Week 7 | -23.2 (37.03) | -22.9 (52.41) | -42.4 (8.45) | -61.6 (10.55) | -44.6 (30.62) |  | -82.4 (20.44) | -27.3 (44.90) | -52.0 (8.41) | -19.4 (11.96)
  Change at Week 8 | -19.5 (40.74) | -29.9 (57.65) | -43.4 (8.98) | -60.7 (11.22) | -44.6 (30.62) |  | -87.3 (14.69) | -37.0 (32.27) | -59.5 (8.96) | -23.1 (12.75)
  Change at Week 9: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 9 | -28.7 (15.95) | 66.0 (22.57) | -42.2 (8.76) | -66.6 (10.13) | -66.9 (0.00) |  | -86.2 (15.97) | -37.3 (35.08) | -63.6 (9.13) | -25.5 (12.99)
  Change at Week 10: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 10 | -21.5 (41.87) | -50.1 (59.26) | -37.4 (8.65) | -76.4 (10.00) | -66.9 (0.00) |  | -88.4 (13.41) | -31.9 (29.47) | -65.9 (9.22) | -25.1 (13.11)
  Change at Week 11: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 11 | -29.0 (31.17) | -49.4 (44.11) | -37.1 (9.54) | -76.5 (11.03) | -66.9 (0.00) |  | -88.4 (13.41) | -35.1 (29.47) | -61.1 (9.12) | -26.1 (12.97)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 12 | -29.3 (34.97) | -49.7 (49.49) | -30.9 (11.35) | -70.1 (13.12) | -66.9 (0.00) |  | -88.4 (13.41) | -33.5 (29.47) | -60.2 (9.58) | -27.0 (13.63)
  Change at Week 13: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 13 | -24.0 (35.58) | -49.7 (50.36) | -35.9 (10.59) | -74.7 (12.24) | -72.8 (0.00) |  | -87.3 (14.69) | -22.7 (32.27) | -63.9 (9.92) | -28.4 (14.11)
  Change at Week 14: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 14 | -20.4 (42.00) | -50.3 (59.44) | -38.2 (9.62) | -71.9 (11.12) | -73.8 (0.00) |  | -85.7 (16.60) | -24.8 (36.48) | -64.9 (9.77) | -29.3 (13.90)
  Change at Week 15: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 15 | -25.9 (37.20) | -49.9 (52.64) | -38.6 (9.08) | -69.7 (10.50) | -73.8 (0.00) |  | -87.9 (14.05) | -27.3 (30.87) | -63.9 (10.34) | -31.3 (14.70)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 16 | -33.5 (35.42) | -49.7 (50.13) | -44.1 (10.40) | -64.0 (12.02) | -73.8 (0.00) |  | -89.0 (12.77) | -19.1 (28.06) | -63.6 (10.16) | -29.4 (14.45)
  Change at Week 17: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 17 | -48.6 (28.92) | -49.0 (40.94) | -41.3 (9.88) | -65.1 (11.42) | -73.8 (0.00) |  | -88.4 (13.41) | -19.2 (29.47) | -58.7 (12.22) | -34.8 (17.38)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 7
  Change at Week 18 | -41.8 (31.93) | -49.4 (45.20) | -42.8 (10.42) | -64.7 (12.04) | -74.7 (0.00) |  | -88.4 (13.41) | -17.6 (29.47) | -58.7 (12.25) | -34.7 (17.43)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 1; Test type: Superiority; p = 0.6532, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 27.7, 80% CI 2-sided [-63.60 to 119.06], Standard Error of Mean 55.77
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 1; Test type: Superiority; p = 0.0187, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 23.6, 80% CI 2-sided [11.38 to 35.85], Standard Error of Mean 9.23
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 1; Test type: Superiority; p = 0.4707, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -39.3, 80% CI 2-sided [-123.27 to 44.68], Standard Error of Mean 44.53
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 1; Test type: Superiority; p = 0.7108, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -1.8, 80% CI 2-sided [-8.22 to 4.59], Standard Error of Mean 4.81
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 2; Test type: Superiority; p = 0.7355, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 22.4, 80% CI 2-sided [-76.47 to 121.23], Standard Error of Mean 60.36
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 2; Test type: Superiority; p = 0.2167, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 16.9, 80% CI 2-sided [-0.66 to 34.52], Standard Error of Mean 13.27
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 2; Test type: Superiority; p = 0.4058, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -63.5, 80% CI 2-sided [-178.16 to 51.13], Standard Error of Mean 60.80
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 2; Test type: Superiority; p = 0.3323, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -6.4, 80% CI 2-sided [-14.95 to 2.15], Standard Error of Mean 6.43
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 3; Test type: Superiority; p = 0.6496, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 34.3, 80% CI 2-sided [-77.29 to 145.80], Standard Error of Mean 68.11
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 3; Test type: Superiority; p = 0.2925, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 13.8, 80% CI 2-sided [-3.12 to 30.70], Standard Error of Mean 12.76
Statistical Analysis 11: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 3; Test type: Superiority; p = 0.4074, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -70.7, 80% CI 2-sided [-198.92 to 57.46], Standard Error of Mean 67.98
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 3; Test type: Other; p = 0.1584, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -15.5, 80% CI 2-sided [-29.60 to -1.49], Standard Error of Mean 10.56
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.7013, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -22.8, 80% CI 2-sided [-111.31 to 65.69], Standard Error of Mean 54.04
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.4230, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 13.4, 80% CI 2-sided [-8.30 to 35.05], Standard Error of Mean 16.35
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.4055, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -60.6, 80% CI 2-sided [-169.90 to 48.69], Standard Error of Mean 57.96
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0709, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -22.7, 80% CI 2-sided [-38.41 to -6.96], Standard Error of Mean 11.82
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 5; Test type: Superiority; p = 0.8268, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 17.7, 80% CI 2-sided [-103.77 to 139.17], Standard Error of Mean 74.17
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 5; Test type: Superiority; p = 0.4082, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 12.4, 80% CI 2-sided [-7.03 to 31.75], Standard Error of Mean 14.63
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 5; Test type: Superiority; p = 0.4818, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -50.4, 80% CI 2-sided [-161.43 to 60.56], Standard Error of Mean 58.86
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 5; Test type: Superiority; p = 0.0673, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -27.1, 80% CI 2-sided [-45.64 to -8.58], Standard Error of Mean 13.93
Statistical Analysis 21: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 6; Test type: Superiority; p = 0.7429, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 29.6, 80% CI 2-sided [-105.00 to 164.10], Standard Error of Mean 82.15
Statistical Analysis 22: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 6; Test type: Superiority; p = 0.1227, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 21.8, 80% CI 2-sided [3.88 to 39.79], Standard Error of Mean 13.55
Statistical Analysis 23: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 6; Test type: Superiority; p = 0.4996, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -47.5, 80% CI 2-sided [-156.95 to 62.02], Standard Error of Mean 58.06
Statistical Analysis 24: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 6; Test type: Superiority; p = 0.0244, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -33.6, 80% CI 2-sided [-51.87 to -15.43], Standard Error of Mean 13.69
Statistical Analysis 25: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 7; Test type: Superiority; p = 0.9967, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -0.3, 80% CI 2-sided [-105.50 to 104.92], Standard Error of Mean 64.24
Statistical Analysis 26: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 7; Test type: Superiority; p = 0.1739, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 19.1, 80% CI 2-sided [1.15 to 37.12], Standard Error of Mean 13.57
Statistical Analysis 27: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 7; Test type: Superiority; p = 0.3978, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -55.1, 80% CI 2-sided [-152.39 to 42.26], Standard Error of Mean 51.61
Statistical Analysis 28: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 7; Test type: Superiority; p = 0.0397, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -32.7, 80% CI 2-sided [-52.26 to -13.07], Standard Error of Mean 14.73
Statistical Analysis 29: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.8922, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 10.4, 80% CI 2-sided [-105.32 to 126.14], Standard Error of Mean 70.66
Statistical Analysis 30: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.2439, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 17.3, 80% CI 2-sided [-1.80 to 36.45], Standard Error of Mean 14.43
Statistical Analysis 31: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.3076, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -50.3, 80% CI 2-sided [-120.29 to 19.61], Standard Error of Mean 37.10
Statistical Analysis 32: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0322, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -36.4, 80% CI 2-sided [-57.32 to -15.55], Standard Error of Mean 15.70
Statistical Analysis 33: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 9; Test type: Superiority; p = 0.0418, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -94.7, 80% CI 2-sided [-139.98 to -49.36], Standard Error of Mean 27.67
Statistical Analysis 34: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 9; Test type: Superiority; p = 0.0865, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 24.4, 80% CI 2-sided [6.49 to 42.26], Standard Error of Mean 13.44
Statistical Analysis 35: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 9; Test type: Superiority; p = 0.3489, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -48.9, 80% CI 2-sided [-124.96 to 27.11], Standard Error of Mean 40.32
Statistical Analysis 36: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 9; Test type: Superiority; p = 0.0286, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -38.1, 80% CI 2-sided [-59.34 to -16.79], Standard Error of Mean 15.99
Statistical Analysis 37: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 10; Test type: Superiority; p = 0.7198, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 28.6, 80% CI 2-sided [-90.32 to 147.59], Standard Error of Mean 72.63
Statistical Analysis 38: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 10; Test type: Superiority; p = 0.0088, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 39.0, 80% CI 2-sided [21.32 to 56.63], Standard Error of Mean 13.27
Statistical Analysis 39: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 10; Test type: Superiority; p = 0.2371, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -56.5, 80% CI 2-sided [-120.39 to 7.34], Standard Error of Mean 33.87
Statistical Analysis 40: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 10; Test type: Superiority; p = 0.0210, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -40.8, 80% CI 2-sided [-62.30 to -19.35], Standard Error of Mean 16.14
Statistical Analysis 41: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 11; Test type: Superiority; p = 0.7312, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 20.4, 80% CI 2-sided [-68.17 to 108.94], Standard Error of Mean 54.07
Statistical Analysis 42: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 11; Test type: Superiority; p = 0.0150, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 39.4, 80% CI 2-sided [19.88 to 58.83], Standard Error of Mean 14.64
Statistical Analysis 43: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 11; Test type: Superiority; p = 0.2559, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -53.3, 80% CI 2-sided [-117.22 to 10.52], Standard Error of Mean 33.87
Statistical Analysis 44: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 11; Test type: Superiority; p = 0.0419, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -35.0, 80% CI 2-sided [-56.21 to -13.72], Standard Error of Mean 15.97
Statistical Analysis 45: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.7589, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 20.4, 80% CI 2-sided [-78.95 to 119.74], Standard Error of Mean 60.66
Statistical Analysis 46: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.0374, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 39.1, 80% CI 2-sided [15.97 to 62.31], Standard Error of Mean 17.42
Statistical Analysis 47: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 12; Test type: Superiority; p = 0.2463, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -54.9, 80% CI 2-sided [-118.80 to 8.93], Standard Error of Mean 33.87
Statistical Analysis 48: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.0632, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -33.2, 80% CI 2-sided [-55.56 to -10.90], Standard Error of Mean 16.78
Statistical Analysis 49: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 13; Test type: Superiority; p = 0.7053, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 25.7, 80% CI 2-sided [-75.41 to 126.78], Standard Error of Mean 61.73
Statistical Analysis 50: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 13; Test type: Superiority; p = 0.0285, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 38.7, 80% CI 2-sided [17.09 to 60.34], Standard Error of Mean 16.25
Statistical Analysis 51: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 13; Test type: Superiority; p = 0.2236, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -64.6, 80% CI 2-sided [-134.58 to 5.32], Standard Error of Mean 37.10
Statistical Analysis 52: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 13; Test type: Other; p = 0.0558, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -35.5, 80% CI 2-sided [-58.65 to -12.41], Standard Error of Mean 17.38
Statistical Analysis 53: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 14; Test type: Superiority; p = 0.7089, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 29.9, 80% CI 2-sided [-89.41 to 149.24], Standard Error of Mean 72.86
Statistical Analysis 54: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 14; Test type: Superiority; p = 0.0347, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 33.7, 80% CI 2-sided [14.08 to 53.35], Standard Error of Mean 14.76
Statistical Analysis 55: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 14; Test type: Superiority; p = 0.2835, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -60.9, 80% CI 2-sided [-139.99 to 18.16], Standard Error of Mean 41.94
Statistical Analysis 56: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 14; Test type: Superiority; p = 0.0525, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -35.5, 80% CI 2-sided [-58.31 to -12.77], Standard Error of Mean 17.11
Statistical Analysis 57: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 15; Test type: Superiority; p = 0.7347, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 24.0, 80% CI 2-sided [-81.68 to 129.66], Standard Error of Mean 64.52
Statistical Analysis 58: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 15; Test type: Superiority; p = 0.0390, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 31.0, 80% CI 2-sided [12.50 to 49.60], Standard Error of Mean 13.94
Statistical Analysis 59: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 15; Test type: Superiority; p = 0.2299, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -60.6, 80% CI 2-sided [-127.49 to 6.33], Standard Error of Mean 35.48
Statistical Analysis 60: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 15; Test type: Superiority; p = 0.0884, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -32.6, 80% CI 2-sided [-56.70 to -8.53], Standard Error of Mean 18.11
Statistical Analysis 61: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.8085, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 16.3, 80% CI 2-sided [-84.37 to 116.87], Standard Error of Mean 61.44
Statistical Analysis 62: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.2283, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 19.9, 80% CI 2-sided [-1.33 to 41.14], Standard Error of Mean 15.96
Statistical Analysis 63: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.1625, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -69.9, 80% CI 2-sided [-130.76 to -9.11], Standard Error of Mean 32.26
Statistical Analysis 64: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.0707, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -34.2, 80% CI 2-sided [-57.87 to -10.52], Standard Error of Mean 17.80
Statistical Analysis 65: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 17; Test type: Superiority; p = 0.9944, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 0.4, 80% CI 2-sided [-81.79 to 82.55], Standard Error of Mean 50.17
Statistical Analysis 66: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 17; Test type: Superiority; p = 0.1327, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 23.9, 80% CI 2-sided [3.71 to 44.05], Standard Error of Mean 15.16
Statistical Analysis 67: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 17; Test type: Superiority; p = 0.1777, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -69.2, 80% CI 2-sided [-133.09 to -5.35], Standard Error of Mean 33.87
Statistical Analysis 68: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 17; Test type: Superiority; p = 0.2796, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -23.9, 80% CI 2-sided [-52.34 to 4.61], Standard Error of Mean 21.40
Statistical Analysis 69: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.8999, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 7.6, 80% CI 2-sided [-83.15 to 98.30], Standard Error of Mean 55.40
Statistical Analysis 70: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Superiority; p = 0.1867, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = 22.0, 80% CI 2-sided [0.68 to 43.23], Standard Error of Mean 15.99
Statistical Analysis 71: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.1717, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -70.8, 80% CI 2-sided [-134.68 to -6.94], Standard Error of Mean 33.87
Statistical Analysis 72: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Superiority; p = 0.2792, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -23.9, 80% CI 2-sided [-52.50 to 4.61], Standard Error of Mean 21.46

17. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score Over Time
Description: The DLQI is a 10-question questionnaire that considers symptoms and feelings, daily activities, leisure, school, personal relationships, and treatment. Each question, except question 7, is answered on a scale of 0 to 3 (0 for not at all, 1 for a little, 2 for a lot, and 3 for very much), taking into account the previous week. For question 7: participants were asked "Over the last week, has your skin prevented you from working or studying?" If answered yes, score=3; If no, a second question will be asked: "Over the last week how much has your skin been a problem at work or studying?" If further answered a lot, score=2; if a little, score=1; if not at all or not relevant, score=0. The DLQI total score is defined as the sum of all 10-question scores with minimum of 0 meaning no effect on quality of life and 30 meaning extremely large effect.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
score on a scale
  Change at Week 4 | -5.8 (1.49) | 0.0 (0.00) | -3.4 (0.86) | -8.0 (1.96) | -4.7 (2.60) |  | -4.5 (2.99) | 0.0 (NA) — 1 participant in this cohort. | -10.0 (1.83) | -0.6 (3.12)
  Change at Week 8 | -6.5 (1.04) | 0.0 (0.00) | -3.6 (1.37) | -8.3 (2.01) | -4.7 (2.60) |  | -3.0 (4.55) | -12.0 (NA) — 1 participant in this cohort. | -11.2 (1.75) | -1.4 (3.33)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -6.5 (1.04) | 0.0 (0.00) | -4.3 (1.53) | -8.3 (2.01) | -7.0 (2.00) |  | -3.0 (4.55) | -12.0 (NA) — 1 participant in this cohort. | -10.7 (1.69) | -1.5 (3.76)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -7.3 (1.55) | 0.0 (0.00) | -4.8 (1.83) | -7.9 (2.25) | -10.0 (1.00) |  | -6.3 (2.29) | -5.0 (NA) — 1 participant in this cohort. | -10.0 (1.82) | -9.5 (2.46)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -6.0 (1.73) | 0.0 (0.00) | -4.4 (2.02) | -8.7 (2.28) | -17.5 (5.50) |  | -6.5 (2.18) | -8.0 (NA) — 1 participant in this cohort. | -9.9 (2.01) | -9.2 (2.04)

18. Secondary Outcome: Percent Change From Baseline in DLQI Total Score Over Time
Description: as for outcome 17
Time Frame: Baseline, Weeks 4, 8, 12, 16, 18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 4 | -51.0 (17.71) | -3.7 (25.35) | -32.8 (8.77) | -52.4 (10.95) | -24.2 (17.01) |  | -53.5 (33.55) | 6.1 (94.72) | -68.2 (11.77) | 4.1 (16.65)
  Change at Week 8 | -54.5 (12.95) | -2.4 (18.53) | -41.1 (13.32) | -56.0 (16.63) | -24.2 (17.01) |  | -32.5 (64.55) | -85.7 (182.21) | -72.2 (10.71) | -2.3 (15.15)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -54.5 (12.95) | -2.4 (18.53) | -48.1 (14.36) | -55.7 (16.59) | -36.4 (0.00) |  | -32.5 (64.55) | -85.7 (182.21) | -72.9 (11.58) | -5.4 (17.75)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -60.5 (15.08) | -2.5 (21.57) | -51.0 (11.94) | -54.0 (13.79) | -61.4 (0.00) |  | -71.9 (23.07) | -41.5 (65.13) | -69.6 (8.18) | -60.7 (12.54)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -52.5 (18.16) | -3.4 (25.99) | -44.0 (12.37) | -61.3 (14.29) | -89.7 (0.00) |  | -75.0 (19.53) | -52.4 (55.14) | -68.7 (9.18) | -62.6 (14.08)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.2289, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -47.3, 80% CI 2-sided [-98.77 to 4.10], Standard Error of Mean 31.41
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.1788, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 19.6, 80% CI 2-sided [0.96 to 38.27], Standard Error of Mean 14.08
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.6544, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -59.6, 80% CI 2-sided [-275.19 to 156.06], Standard Error of Mean 114.35
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0023, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -72.2, 80% CI 2-sided [-99.39 to -45.09], Standard Error of Mean 20.40
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.1081, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -52.1, 80% CI 2-sided [-89.68 to -14.47], Standard Error of Mean 22.96
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.4926, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 14.9, 80% CI 2-sided [-13.39 to 43.26], Standard Error of Mean 21.37
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.8315, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 53.2, 80% CI 2-sided [-361.63 to 467.98], Standard Error of Mean 219.98
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0014, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -69.9, 80% CI 2-sided [-94.61 to -45.22], Standard Error of Mean 18.56
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.1081, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -52.1, 80% CI 2-sided [-89.68 to -14.47], Standard Error of Mean 22.96
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.7339, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 7.6, 80% CI 2-sided [-21.65 to 36.82], Standard Error of Mean 21.97
Statistical Analysis 11: Comparison: Placebo: LSC Cohort vs KPL-716: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.8315, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 53.2, 80% CI 2-sided [-361.63 to 467.98], Standard Error of Mean 219.98
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.0055, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -67.6, 80% CI 2-sided [-95.92 to -39.22], Standard Error of Mean 21.26
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.1188, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -57.9, 80% CI 2-sided [-101.70 to -14.15], Standard Error of Mean 26.73
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.8697, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 3.0, 80% CI 2-sided [-21.26 to 27.35], Standard Error of Mean 18.27
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.7368, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -30.3, 80% CI 2-sided [-178.62 to 117.94], Standard Error of Mean 78.64
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.5571, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -9.0, 80% CI 2-sided [-29.03 to 11.03], Standard Error of Mean 15.02
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.2251, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -49.1, 80% CI 2-sided [-101.80 to 3.69], Standard Error of Mean 32.21
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Superiority; p = 0.3733, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 17.3, 80% CI 2-sided [-7.90 to 42.48], Standard Error of Mean 18.93
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.7662, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -22.6, 80% CI 2-sided [-148.16 to 102.89], Standard Error of Mean 66.57
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Other; p = 0.7241, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -6.1, 80% CI 2-sided [-28.54 to 16.44], Standard Error of Mean 16.87

19. Secondary Outcome: Change From Baseline in ItchyQoL Total Score Over Time
Description: ItchyQoL focuses on impact of pruritus on daily activities and on the level of psychological stress. It contains 22 items. The frequency items are scored using a 5-point Likert scale ranging from "never" to "all the time". The bother items are scored from 1 (not bothered) to 5 (severely bothered). The recall period in ItchyQoL is the past week. The ItchyQoL total score is defined as the sum of all 22-items scores. Total scores can be classified as little (0-30), mild (31-50), moderate (51-80), and severe (81-110).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 18
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
score on a scale
  Change at Week 4 | -17.0 (13.07) | 0.0 (0.00) | -10.9 (3.63) | -18.9 (6.25) | -27.3 (15.32) |  | -31.5 (13.91) | 0.0 (NA) — 1 participant in this cohort. | -29.0 (5.61) | -16.9 (7.04)
  Change at Week 8 | -23.3 (9.08) | -0.5 (0.50) | -17.8 (4.61) | -20.8 (8.66) | -27.3 (15.32) |  | -38.8 (15.84) | -10.0 (NA) — 1 participant in this cohort. | -35.8 (5.88) | -23.1 (7.31)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -22.8 (11.74) | 0.0 (0.00) | -22.0 (5.96) | -19.2 (5.78) | -47.0 (6.00) |  | -41.5 (11.99) | -18.0 (NA) — 1 participant in this cohort. | -35.5 (6.54) | -27.3 (4.62)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -33.3 (11.46) | 0.0 (0.00) | -19.9 (5.18) | -18.1 (6.93) | -50.0 (3.00) |  | -41.5 (11.89) | -18.0 (NA) — 1 participant in this cohort. | -38.1 (5.66) | -29.2 (8.15)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -29.3 (9.68) | 0.0 (0.00) | -25.1 (7.18) | -21.4 (6.82) | -64.5 (14.50) |  | -46.8 (8.62) | -15.0 (NA) — 1 participant in this cohort. | -32.9 (6.40) | -31.8 (8.46)

20. Secondary Outcome: Percent Change From Baseline in ItchyQoL Total Score Over Time
Description: as for outcome 19
Time Frame: Baseline, Weeks 4, 8, 12, 16, 18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change
  Change at Week 4 | -21.4 (16.56) | -0.2 (23.57) | -13.0 (5.15) | -24.3 (6.43) | -29.1 (7.02) |  | -47.8 (17.37) | 39.7 (46.22) | -34.8 (5.84) | -14.6 (8.32)
  Change at Week 8 | -29.2 (11.47) | -0.6 (16.32) | -23.7 (7.21) | -26.0 (9.01) | -29.1 (7.02) |  | -56.3 (23.23) | 27.3 (61.79) | -42.7 (6.29) | -21.9 (8.97)
  Change at Week 12: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 12 | -28.3 (14.70) | 0.2 (20.91) | -29.4 (6.30) | -25.0 (7.29) | -50.9 (0.00) |  | -58.2 (15.85) | 12.0 (42.18) | -42.7 (6.58) | -26.0 (10.25)
  Change at Week 16: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 16 | -41.7 (14.66) | -0.2 (20.86) | -26.5 (6.61) | -23.2 (7.65) | -54.6 (0.00) |  | -59.8 (12.34) | 19.8 (32.82) | -45.8 (6.06) | -29.4 (9.44)
  Change at Week 18: number analyzed (Participants) | 4 | 2 | 12 | 9 | 2 | 0 | 4 | 1 | 14 | 6
  Change at Week 18 | -36.6 (12.16) | 0.0 (17.30) | -32.5 (7.93) | -27.6 (9.17) | -69.2 (0.00) |  | -63.8 (7.49) | 10.2 (19.94) | -39.6 (7.06) | -31.7 (11.00)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 4; Test type: Superiority; p = 0.5195, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -21.1, 80% CI 2-sided [-68.69 to 26.43], Standard Error of Mean 29.04
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 4; Test type: Superiority; p = 0.1869, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 11.3, 80% CI 2-sided [0.34 to 22.26], Standard Error of Mean 8.27
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 4; Test type: Superiority; p = 0.2545, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -87.5, 80% CI 2-sided [-191.75 to 16.79], Standard Error of Mean 55.30
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 4; Test type: Superiority; p = 0.0643, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -20.2, 80% CI 2-sided [-33.88 to -6.57], Standard Error of Mean 10.26
Statistical Analysis 5: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 8; Test type: Superiority; p = 0.2503, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -28.6, 80% CI 2-sided [-61.52 to 4.35], Standard Error of Mean 20.11
Statistical Analysis 6: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 8; Test type: Superiority; p = 0.8468, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = 2.3, 80% CI 2-sided [-13.08 to 17.62], Standard Error of Mean 11.58
Statistical Analysis 7: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 8; Test type: Superiority; p = 0.3755, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -83.6, 80% CI 2-sided [-222.98 to 55.18], Standard Error of Mean 73.93
Statistical Analysis 8: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 8; Test type: Superiority; p = 0.0755, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -20.9, 80% CI 2-sided [-35.58 to -6.15], Standard Error of Mean 11.06
Statistical Analysis 9: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 12; Test type: Superiority; p = 0.3486, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -28.6, 80% CI 2-sided [-70.76 to 13.65], Standard Error of Mean 25.77
Statistical Analysis 10: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 12; Test type: Superiority; p = 0.6559, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -4.4, 80% CI 2-sided [-17.28 to 8.50], Standard Error of Mean 9.69
Statistical Analysis 11: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 12; Test type: Superiority; p = 0.2987, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -70.2, 80% CI 2-sided [-165.35 to 24.94], Standard Error of Mean 50.46
Statistical Analysis 12: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 12; Test type: Superiority; p = 0.1966, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -16.7, 80% CI 2-sided [-33.29 to -0.13], Standard Error of Mean 12.43
Statistical Analysis 13: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 16; Test type: Superiority; p = 0.2051, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -41.5, 80% CI 2-sided [-83.56 to 0.62], Standard Error of Mean 25.70
Statistical Analysis 14: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 16; Test type: Superiority; p = 0.7511, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -3.3, 80% CI 2-sided [-16.79 to 10.25], Standard Error of Mean 10.16
Statistical Analysis 15: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 16; Test type: Superiority; p = 0.1797, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -79.6, 80% CI 2-sided [-153.68 to -5.59], Standard Deviation 39.27
Statistical Analysis 16: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 16; Test type: Superiority; p = 0.1715, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -16.3, 80% CI 2-sided [-31.61 to -1.08], Standard Error of Mean 11.45
Statistical Analysis 17: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Change at Week 18; Test type: Superiority; p = 0.1850, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -36.5, 80% CI 2-sided [-71.47 to -1.63], Standard Error of Mean 21.32
Statistical Analysis 18: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Change at Week 18; Test type: Superiority; p = 0.6907, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -4.9, 80% CI 2-sided [-21.15 to 11.29], Standard Error of Mean 12.19
Statistical Analysis 19: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Change at Week 18; Test type: Superiority; p = 0.0901, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -74.0, 80% CI 2-sided [-118.97 to -29.02], Standard Error of Mean 23.85
Statistical Analysis 20: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Change at Week 18; Test type: Superiority; p = 0.5640, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS Mean Difference = -7.8, 80% CI 2-sided [-25.64 to 9.94], Standard Error of Mean 13.34

21. Primary Outcome: Percent Change From Baseline in Weekly Average WI-NRS at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | KPL-716: CIU Cohort | Placebo: CIU Cohort | KPL-716: CIP Cohort | Placebo: CIP Cohort | KPL-716: LP Cohort | Placebo: LP Cohort | KPL-716: LSC Cohort | Placebo: LSC Cohort | KPL-716: PPs Cohort | Placebo: PPs Cohort
Number analyzed (Participants) | 4 | 2 | 14 | 9 | 3 | 0 | 4 | 1 | 14 | 7
percent change | -50.7 (21.56) | -19.0 (31.07) | -52.4 (9.32) | -48.8 (11.63) | -39.4 (10.21) |  | -85.0 (11.76) | 7.0 (26.80) | -66.5 (7.78) | -29.0 (11.00)
Statistical Analysis 1: Comparison: KPL-716: CIU Cohort vs Placebo: CIU Cohort; Test type: Superiority; p = 0.4734, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -31.7, 80% CI 2-sided [-95.11 to 31.76], Standard Error of Mean 38.73
Statistical Analysis 2: Comparison: KPL-716: CIP Cohort vs Placebo: CIP Cohort; Test type: Superiority; p = 0.8130, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -3.6, 80% CI 2-sided [-23.33 to 16.18], Standard Error of Mean 14.91
Statistical Analysis 3: Comparison: KPL-716: LSC Cohort vs Placebo: LSC Cohort; Test type: Superiority; p = 0.0979, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -92.0, 80% CI 2-sided [-150.60 to -33.32], Standard Error of Mean 31.10
Statistical Analysis 4: Comparison: KPL-716: PPs Cohort vs Placebo: PPs Cohort; Test type: Superiority; p = 0.0122, ANCOVA — Calculated from an ANCOVA model including treatment as factor and baseline values as covariate; LS mean difference = -37.5, 80% CI 2-sided [-55.48 to -19.61], Standard Error of Mean 13.48

ADVERSE EVENTS:
Time Frame: From first dose of study treatment through the end-of-study visit (Week 18).
Description: The adverse event data are presented by combined cohorts for public reporting purposes because the low numbers of participants in the individual disease-specific cohorts may cause re-identification concerns if presented separately.
Arm/Group | KPL-716 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/39 | 0/19
Other Adverse Events (participants affected / at risk) | 15/39 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KPL-716 (N=39) | Placebo (N=19)
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KPL-716 (N=39) | Placebo (N=19)
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2
Cardiac murmur (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Electrocardioagram T wave abnormal (Investigations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Chalazion (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the first right to publish study results. PI may publish study results after Sponsor publishes the study results or 18 months after study completion at all participating sites, whichever comes first, provided that Sponsor may embargo such publication for up to 60 days for purposes of identifying confidential information that must be removed and up to an additional 60 days to prepare a patent application if there is patentable subject matter in the PI's proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03858634/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03858634/SAP_001.pdf